| | Statistical Arialysis Flati Fillal |
|---|---|
| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
| Detailed Title: | A phase III, open-label, single-group, multi-centre study to assess the immunogenicity, safety and reactogenicity of GSK Biologicals' combined reduced antigen content diphtheria, tetanus and acellular pertussis (dTpa) vaccine, <i>Boostrix</i> , administered as a booster dose in healthy Russian subjects aged four years and older. |
| eTrack study number and<br>Abbreviated Title | 201532 [DTPA (BOOSTRIX)-050] |
| Scope: | All analyses as planned per protocol and for study report. |
| Date of Statistical Analysis<br>Plan | 09-OCT-2017 |
| Co-ordinating author: | (Lead Statistician) |
| Reviewed by: | R&D Project Leader) PPD , Clinical Research and Development Lead (CRDL) PPD (Study statistician) PPD (peer reviewer statistician) PPD (public disclosure) (Scientific writer) PPD (Lead statistical analyst) PPD (Global Regulatory Affairs) Ivonne PPD and PPD (Safety Physician) |
| Approved by: | R&D Project Leader) PPD , Clinical Research and Development Lead (CRDL) PPD (Study statistician) PPD (Lead Statistician) PPD (Lead statistical analyst) PPD (Scientific writer) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 14April 2017)

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| LIS | T OF A | ABBREVIATIONS | 7 |
| 1. | DOC | UMENT HISTORY | 9 |
| 2. | STUE | DY DESIGN | 9 |
| 3. | OR IE | ECTIVES | 10 |
| ٥. | 3.1. | | |
| | 3.2. | | 10 |
| 4. | ENDE | POINTS | 11 |
| т. | 4.1. | | |
| | 4.2. | | |
| 5. | ANAL | LYSIS SETS | 12 |
| | 5.1. | Definition | |
| | | 5.1.1. Total vaccinated cohort (TVC) | 12 |
| | | 5.1.2. Per protocol cohort for analysis of immunogenicity | 12 |
| | 5.2. | Criteria for eliminating data from Analysis Sets | 13 |
| | | 5.2.1. Elimination from Total vaccinated cohort (TVC) | |
| | | 5.2.2. Elimination from ATP cohort for immunogenicity | 14 |
| | | 5.2.2.1. Excluded subjects | |
| | | 5.2.2.2. Right censored Data | |
| | | 5.2.2.3. Visit-specific censored Data | 15 |
| | 5.3. | Important protocol deviation not leading to elimination from ATP cohort for immunogenicity | 15 |
| | | • , | |
| 6. | STAT | FISTICAL ANALYSES | |
| | 6.1. | Demography | |
| | | 6.1.1. Analysis of demographics/baseline characteristics planne | |
| | | in the protocol | |
| | | 6.1.2. Additional considerations | |
| | 6.2. | Exposure | |
| | | 6.2.1. Analysis of exposure planned in the protocol | |
| | | 6.2.2. Additional considerations | |
| | 6.3. | Immunogenicity | |
| | | 6.3.1. Analysis of immunogenicity planned in the protocol | |
| | | 6.3.2. Additional considerations | |
| | 6.4. | Analysis of safety | |
| | | 6.4.1. Analysis of safety planned in the protocol | |
| | | 6.4.2. Additional considerations | 19 |
| 7. | ANAL | LYSIS INTERPRETATION | 20 |
| 8. | CONI | DUCT OF ANALYSES | 20 |
| | 8.1. | Sequence of analyses | |
| | 8.2. | Statistical considerations for interim analyses | 20 |
| | 8.3. | · · | |

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

| 9. | CHAN | GES FRO | OM PLANNED ANALYSES | 20 |
|---|---|---|---|---|
| 10. | LIST ( | OF FINAL | REPORT TABLES, LISTINGS AND FIGUR | RES21 |
| 11. | | _ | NDARD DATA DERIVATION RULE AND S | |
| | | | al Method References | |
| | 11.2. | Standard | d data derivation | 22 |
| | | 11.2.1. | Date derivation | 22 |
| | | | Demography | |
| | | 11.2.3. | Immunogenicity | 22 |
| | | 11.2.4. | Safety | <mark>2</mark> 3 |
| 12. | ANNE | X 2: SUM | IMARY ON ELIMINATION CODES | 27 |
| 13 | ANNF | X 3· STU | DY SPECIFIC MOCK TEL | 27 |

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

## **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Study group and epoch foreseen in the study | 10 |
| Table 2 | Study group and treatment foreseen in the study | 10 |
| Table 3 | Blinding of study epoch | 10 |
| Table 4 | Age stratification | 16 |
| Table 5 | Humoral Immunity (Antibody determination) | 18 |
| Table 6 | Intensity scales to be used by the parent(s)/LAR(s) for solicited symptoms during the solicited follow-up period | 24 |
| Table 7 | Intensity scales for solicited symptoms in adults and children of six years of age or more | 25 |

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

## **LIST OF TEMPLATES**

| | P | AGE |
|---|---|---|
| Template 1 | Number of subjects enrolled by center (Total Vaccinated Cohort) | 28 |
| Template 2 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal at Visit 3 (Total Vaccinated Cohort) | 28 |
| Template 3 | Number of subjects at each visit and list of withdrawn subjects (Total Vaccinated Cohort) | 29 |
| Template 4 | Number of subjects enrolled into the study as well as the number of subjects excluded from ATP analyses with reasons for exclusion | 30 |
| Template 5 | Deviations from specifications for age and intervals between study visits (Total Vaccinated Cohort) | 31 |
| Template 6 | Summary of demographic characteristics (ATP cohort for Immunogenicity) | 31 |
| Template 7 | Summary of vital signs characteristics (Total Vaccinated Cohort) | 32 |
| Template 8 | Study population (Total Vaccinated Cohort) | 32 |
| Template 9 | Seropositivity and seroprotection rates and GMCs for anti-<br>diphtheria and anti-tetanus antibodies before and one month<br>after the booster vaccination (ATP cohort for immunogenicity) | 33 |
| Template 10 | Booster responses for anti-PT, anti-FHA and anti-PRN antibody concentration one month after the booster vaccination (ATP cohort for immunogenicity) | 34 |
| Template 11 | Reverse cumulative curve for anti-diphtheria antibody concentration one month after the booster vaccination (ATP cohort for immunogenicity) | 35 |
| Template 12 | Seroprotection rate for anti-Diphtheria antibody concentration by ELISA and VERO NEUTRALISATION (ATP cohort) | 36 |
| Template 13 | Compliance in returning symptom information (Total Vaccinated Cohort) | 36 |
| Template 14 | Incidence and nature of grade 3 symptoms (solicited and unsolicited) reported during the 4-day (Days 0-3) period after vaccination following each dose and overall (Total Vaccinated Cohort) | 37 |
| Template 15 | Incidence of solicited local symptoms reported during the 4-day (Days 0-3) period after vaccination following each dose and overall (Total Vaccinated Cohort) | 37 |

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

| Template 16 | Incidence of solicited general symptoms reported during the 4-day (Days 0-3) post-vaccination period (Total Vaccinated Cohort). | 38 |
|---|---|---|
| Template 17 | Percentage of subjects with grade 3 unsolicited symptoms classified by MedDRA SOC and PT from Day 0 to Day 30 after any vaccination (Total Vaccinated Cohort) | 39 |
| Template 18 | Number (%) of subjects with serious adverse events from first study vaccination up to Visit 3 including number of events reported (Total Vaccinated Cohort) | 41 |
| Template 19 | Subjects with Serious Adverse Events reported up to Visit 2 (Total Vaccinated Cohort) | 42 |
| Template 20 | Number and percentage of subjects who started at least one concomitant medication from Day 0 to Day 7 (Total Vaccinated Cohort) | 44 |
| Template 21 | Solicited and Unsolicited symptoms experienced by subjects classified by MedDRA Primary System Organ Class and Preferred Term within the 31-day (Days 0-30) post-vaccination period - SAE excluded (Total vaccinated cohort) | 44 |
| Template 22 | Minimum and maximum activity dates (TVC) | 44 |
| Template 23 | Number of enrolled subjects by age category (TVC) | 45 |
| Template 24 | Number of subjects by country | 45 |
| Template 25 | Listing of dropouts due to AEs, SAEs and solicited symptoms (Total cohort) | 45 |
| Template 26 | Percentage of subjects with large injection site reaction during the 4-day (Days 0-3) period after Boostrix (Total Vaccinated Cohort) | 46 |

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

#### LIST OF ABBREVIATIONS

AE Adverse event

ANOVA Analysis of Variance

BS Blood Sample

cDISCI Clinical Data Interchange Standards Consortium

CI Confidence Interval

CRF Case Report Form

CTRS Clinical Trial Registry Summary

EL.U/ml ELISA unit per milliliter

Eli Type Internal GSK database code for type of elimination code

ELISA Enzyme-linked immunosorbent assay

GE Gastroenteritis

GSK GlaxoSmithKline

iDMC Independent Data Monitoring Committee

IU/ml International units per milliliter

LL Lower Limit of the confidence interval

MedDRA Medical Dictionary for Regulatory Activities

N.A. Not Applicable

PD Protocol Deviation

ATP Per Protocol Set

SAE Serious adverse event

SAP Statistical Analysis Plan

SAS Statistical Analysis Software

SBIR GSK Biological's Internet Randomization System

SD Standard Deviation

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

SR Study Report

TFL Tables Figures and Listings

TOC Table of Content

TVC Total Vaccinated Cohort

UL Upper Limit of the confidence interval

### 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|---------------|--------------------------------------|
| 09-Oct-2017 | first version | Amendment 02 Final 1: 07 August 2017 |

#### 2. STUDY DESIGN



<u>Visit:</u> <u>Visit 1</u> <u>Day 1</u> Day 31

**Blood sampling:** Pre-Booster Post-Booster

Vaccination Study End

Age: ≥ 4 yrs

Protocol waivers or exemptions are not allowed unless necessary for the management of immediate safety concerns. Therefore, adherence to the study design requirements, including those specified in the outline of study procedures (Section 5.5 of the protocol), are essential and required for study conduct.

- Experimental design: Phase III, open-label, non-randomised, multi-centric, single-country study with a single group.
- Duration of the study:
  - Epoch 001: Primary Epoch starting at Visit 1 (Day 1) and ending at Visit 2 (Day 31)
- Primary Completion Date (PCD): Visit 2 (Day 31)
- End of Study (EoS): Last testing results released of samples collected at Visit 2.
- Study groups: The study group and epoch foreseen in this study is presented in Table 1.

<sup>\*</sup> An equal number of subjects are expected to be recruited in the following age categories: 4-9 years (children), 10-17 years (adolescents), 18-64 years (adults) and ≥65 years (elderly population) in order to evaluate data.

Table 1 Study group and epoch foreseen in the study

| Study group | Number of subjects | Age (Min) | Epoch |
|-------------|--------------------|-----------|-----------|
| | | | Epoch 001 |
| dTpa Group | 448 | ≥4 years | X |

## Table 2 Study group and treatment foreseen in the study

| Treatment name | Vaccine/Product name | Study Group |
|----------------|----------------------|-------------|
| Treatment name | vaccine/Froduct name | dTpa Group |
| Boostrix | dTpa | X |

- Control: uncontrolled (in terms of no active comparator).
- Vaccination schedule: A single dose of *Boostrix* vaccine will be administered to all subjects at Visit 1 (Day 1).
- Treatment allocation: Non-randomised and stratified by age.
- Blinding: open.

Table 3 Blinding of study epoch

| Study Epoch | Blinding |
|-------------|----------|
| Epoch 001 | open |

- Sampling schedule: A blood sample of approximately 5 ml will be collected from all subjects before vaccination (at the Pre-Booster timepoint) and one month after vaccination (Post-Booster timepoint).
- Type of study: self-contained.
- Data collection: Electronic Case Report Form (eCRF).

#### 3. OBJECTIVES

# 3.1. Primary objectives

• To assess the immune response to the dTpa vaccine in terms of seroprotection status for antibodies against diphtheria and tetanus antigens and in terms of seropositivity status for antibodies against the pertussis antigens [pertussis toxoid (PT), filamentous haemagglutinin (FHA) and pertactin (PRN)], one month after vaccination.

Refer to Section 4.1 for the definition of the primary endpoints.

# 3.2. Secondary objectives

- To assess the immune response in terms of booster response\* to diphtheria, tetanus, PT, FHA, and PRN antigens, one month after vaccination.
- To assess the immune response in terms of antibody concentrations to diphtheria, tetanus, PT, FHA, and PRN antigens, one month after vaccination.

• To assess the reactogenicity and safety of Boostrix in terms of solicited symptoms (local and general), unsolicited adverse events (AEs) and serious adverse events (SAEs).

Refer to Section 4.2 for the definition of the secondary endpoints.

#### 4. ENDPOINTS

## 4.1. Primary endpoints

- Immunogenicity with respect to components of the study vaccine.
  - o Anti-diphtheria\* and anti-tetanus seroprotection status (ie antibody concentrations ≥0.1 IU/ml), one month after vaccination.
  - o Anti-PT, anti-FHA and anti-PRN seropositivity status (ie antibody concentration is greater than or equal to the assay cut-off value), one month after vaccination.

## 4.2. Secondary endpoints

- Booster response to the diphtheria, tetanus and pertussis (PT, FHA and PRN) antigens, one month after vaccination.
  - o Booster response to Diphtheria and Tetanus antigens is defined as:
    - for subjects with pre-vaccination antibody concentration <0.1 IU/ml (i.e. below the seroprotection cut-off), antibody concentrations at least ≥0.4 IU/ml, one month after vaccination, and
    - for subjects with pre-vaccination antibody concentration ≥0.1 IU/ml (i.e. equal or above the seroprotection cut-off), an increase in antibody concentrations of at least four times the pre-vaccination concentration, one month after vaccination.
  - o Booster response to PT, FHA and PRN antigens is defined as:
    - for subjects with pre-vaccination antibody concentration below the assay cut-off, post-vaccination antibody concentration ≥ four times the assay cutoff,
    - for subjects with pre-vaccination antibody concentration between the assay cut-off and below four times the assay cut-off, post-vaccination antibody concentration ≥ four times the pre-vaccination antibody concentration, and
    - for subjects with pre-vaccination antibody concentration ≥ four times the assay cut-off, post-vaccination antibody concentration ≥ two times the pre-vaccination antibody concentration
- Immunogenicity with respect to components of the study vaccine.
  - o Anti-diphtheria anti-tetanus, anti-PT, anti-FHA and anti-PRN antibody concentrations, one month after vaccination.

<sup>\*</sup>Sera with ELISA concentrations <0.1 IU/ml will be tested for neutralising antibodies using a Vero-cell neutralisation assay.

- Solicited local and general symptoms.
  - Occurrence of each solicited local and general symptom during the 4-day (Day 1-4) follow-up period after vaccination.
  - Occurrence of large swelling reactions during the 4-day (Day 1-4) follow-up period after vaccination.
- Unsolicited adverse events.
  - Occurrence of unsolicited AEs during the 31-day (Day 1-31) follow-up period after vaccination, according to the Medical Dictionary for Regulatory Activities (MedDRA) classification.
- Serious adverse events.
  - Occurrence of SAEs from the vaccination up to study end.

#### 5. ANALYSIS SETS

#### 5.1. Definition

#### 5.1.1. Total vaccinated cohort (TVC)

The TVC will include all subjects with at least one study vaccine administration documented.

- A safety analysis based on the TVC will include all vaccinated subjects.
- An immunogenicity analysis based on the TVC will include all vaccinated subjects for whom immunogenicity data are available.

Note that enrolled subjects who gave informed consent or blood sample pre-vaccination but were not vaccinated will be excluded from TVC.

# 5.1.2. Per protocol cohort for analysis of immunogenicity

The PP cohort for immunogenicity will include all evaluable subjects:

- Who have received the dose of study vaccine.
- For whom administration site of study vaccine is known and according to the protocol.
- Who have not received a vaccine not specified or forbidden in the protocol.
- Who meet all eligibility criteria.
- Who are within the maximum interval (the interval between Visit 1 and blood sampling at Visit 2, considered for inclusion of a subject will be 21–48 days) allowed as defined in the protocol.

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

- Who did not receive a product leading to exclusion from a PP analysis (refer to Section 6.7.2 of the protocol, namely
  - Any investigational or non-registered product (drug or vaccine) other than the study vaccine used during the study period.
  - o Immunosuppressants or other immune-modifying drugs administered chronically (i.e. more than 14 days) during the study period. For corticosteroids, this will mean prednisone ≥20 mg/day (for adult subjects) or ≥0.5 mg/kg/day (for paediatric subjects), or equivalent. Inhaled and topical steroids are allowed.
  - o Long-acting immune-modifying drugs administered at any time during the study period (e.g. infliximab).
  - A vaccine not foreseen by the study protocol administered during the period starting from the dose of study vaccine (Day 1) and ending 31 days after the dose of vaccine administration, with the exception of influenza vaccine which is allowed throughout the study period.
  - In case an emergency mass vaccination for an unforeseen public health threat (e.g.: a pandemic) is organised by the public health authorities, outside the routine immunisation program, the time period described above can be reduced if necessary for that vaccine provided it is licensed and used according to its Summary of Product Characteristics (SmPC) and according to the local governmental recommendations and provided a written approval of the Sponsor is obtained
  - Immunoglobulins and/or any blood products administered during the study period.)
- Who did not present with a medical condition leading to exclusion from an PP analysis (refer to Section 6.8 of the protocol, namely subjects will be eliminated from the PP cohort for immunogenicity if, during the study, they incur a condition that has the capability of altering their immune response or are confirmed to have an alteration of their initial immune status).
- For whom data concerning immunogenicity endpoint measures are available post vaccination. This will include subjects for whom assay results are available for antibodies against at least one study vaccine antigen component.

# 5.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each sets.

## 5.2.1. Elimination from Total vaccinated cohort (TVC)

Code 1030 (Study vaccine not administered at all) and code 900 (invalid informed consent or fraud data) will be used for identifying subjects eliminated from TVC.

# 5.2.2. Elimination from ATP cohort for immunogenicity

# 5.2.2.1. Excluded subjects

A subject will be excluded from the ATP cohort for immunogenicity under the following conditions

| Code | Decode => Condition under which the code is used |
|---|---|
| 900 | Questionable subject => Invalid informed consent or fraudulent data. In case informed consent is obtained retrospectively the subject is not eliminated. |
| 1030 | Study vaccine dose not administrated at all but subject number allocated => subjects enrolled but not vaccinated |
| 1040 | Administration of vaccine(s) forbidden in the protocol => O Any investigational or non-registered product (drug or vaccine) other than the study vaccine used during the study period. |
| | O A vaccine not foreseen by the study protocol administered during the period starting from the dose of study vaccine (Day 1) and ending 31 days after the dose of vaccine administration, with the exception of influenza vaccine which is allowed throughout the study period. This includes emergency mass vaccination for an unforeseen public health threat (e.g.: a pandemic) organised by the public health authorities, outside the routine immunisation program. |
| 1070 | Study vaccine dose not administered according to protocol => for instance • Route of vaccination is not Intramuscular for Boostrix |
| | Wrong reconstitution of Boostrix before injection |
| 1080 | Vaccine temperature deviation => Boostrix vaccine administered despite a Good Manufacturing Practices (GMP) no-go temperature deviation |
| 1090 | Expired vaccine administered=> Subjects who received an expired Boostrix vaccine |
| 2010 | Protocol violation (inclusion/exclusion criteria) => ineligible subject: • age below (excluding) 4 year |
| | <ul> <li>Other considerations as stated in section 4.2 – 4.3 in the protocol</li> </ul> |

| | Statistical Arialysis Frant Final |
|---|---|
| 2040 | Administration of any medication forbidden by the protocol=> |
| | <ul> <li>Immunosuppressants or other immune-modifying drugs<br/>administered chronically (i.e. more than 14 days) during the<br/>study period. For corticosteroids, this will mean prednisone<br/>≥20 mg/day (for adult subjects) or ≥0.5 mg/kg/day (for<br/>paediatric subjects), or equivalent. Inhaled and topical steroids<br/>are allowed.</li> </ul> |
| | <ul> <li>Long-acting immune-modifying drugs administered at any<br/>time during the study period (e.g. infliximab).</li> </ul> |
| | <ul> <li>Immunoglobulins and/or any blood products administered<br/>during the study period.)</li> </ul> |
| 2070 | Concomitant infection not related to the vaccine which may influence immune response = > subject who incurs a condition that has the capability of altering their immune response or are confirmed to have an alteration of their initial immune status |
| 2090 | Non-compliance with the blood sampling schedule (including wrong and unknown dates) => Blood sample not collected within 21 days-48 days after the Boostrix vaccine. |
| 2100 | Essential serological data missing => No serological results at all available post-vaccination (Visit 2) |
| 2120 | Obvious incoherence or abnormality or error in data => BS result available while BS not taken |
| | <ul> <li>Post vaccination results below pre-vaccination results for all<br/>available assays tested at pre-vaccination ie PT, FHA, PRN,<br/>Diphtheria (ELISA), Tetanus</li> </ul> |

### 5.2.2.2. Right censored Data

Not applicable

## 5.2.2.3. Visit-specific censored Data

Not applicable

# 5.3. Important protocol deviation not leading to elimination from ATP cohort for immunogenicity

Refer to the protocol deviaito management plan for important protocol deviation not leading to elimination from ATP cohort for immunogenicity.

#### 6. STATISTICAL ANALYSES

Note that standard data derivation rule and stat methods are described in annex 1 and will not be repeated below.

## 6.1. Demography

# 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

Demographic characteristics (age at vaccination visit in years, gender and geographical ancestry, body mass index in kg/m<sup>2</sup>), cohort description and withdrawal status will be summarised using descriptive statistics:

- Frequency tables will be generated for categorical variable such as centre.
- Mean, median, standard deviation will be provided for continuous data such as age.
- The distribution of subjects based on age stratification will be tabulated (as seen in Table 4).

In addition, the above analysis will also be done for sub-groups based on age as an exploratory analysis.

Table 4 Age stratification

| Age groups | Number of subjects |
|-------------|--------------------|
| 4-9 years | ~112 |
| 10-17 years | ~112 |
| 18-64 years | ~112 |
| ≥65 years | ~112 |

#### 6.1.2. Additional considerations

All demography summaries will be generated for the TVC and ATP cohort. An additional age split will be added in the 4-9 years group to determine the distribution of subjects below 6 year old as solicited symptoms are different (see section 11.2.4).

Number and reason for elimination from ATP will be tabulated.

## 6.2. Exposure

## 6.2.1. Analysis of exposure planned in the protocol

Not described in the protocol as a single dose is provided and the number of vaccinated subjects is provided.

#### 6.2.2. Additional considerations

Not applicable.

## 6.3. Immunogenicity

## 6.3.1. Analysis of immunogenicity planned in the protocol

The primary analysis will be based on the PP cohort for analysis of immunogenicity. If, the percentage of vaccinated subjects with serological results excluded from the PP cohort for analysis of immunogenicity is 5% or more, a second analysis based on the TVC will be performed to complement the PP analysis.

For all subjects and each antigen:

- Seropositivity/seroprotection rate at pre-vaccination and one month post-vaccination will be calculated with exact 95% CIs.
- GMCs at pre-vaccination and one month post-vaccination will be tabulated with 95% CIs.
- Booster response rate one month post-vaccination will be calculated with exact 95% CIs for diphtheria, tetanus and pertussis antigens.

In addition, the above analysis will also be done based on age stratification (Refer Table 4) as an exploratory analysis.

Finally, antibody concentrations distribution at pre-vaccination and one month post-vaccination will be displayed using reverse cumulative curves (RCC).

## Handling of missing data:

• For a given subject and a given immunogenicity measurement, missing or non-evaluable measurements will not be replaced. Therefore, an analysis will exclude subjects with missing or non-evaluable measurements.

#### 6.3.2. Additional considerations

Seroprotection and booster response is defined in section 4. The percentage of subjects with ELISA anti-Diphtheria above 0.1 IU/ml or with Vero anti-Diphtheria above 0.01 IU/ml will be summarized at pre and post vaccination. In case subjects with ELISA anti-Diphtheria above 0.1 IU/ml have no result by Vero, the subjects will be treated as censored for Vero anti-Diphtheria and survival method will be used to estimate percentage and associated CI.

A seronegative subject is a subject whose antibody concentration is below the assay cutoff value. A seropositive subject is a subject whose antibody concentration is greater than or equal to the assay cut-off value.

The thresholds defining seropositivity are provided below

Table 5 Humoral Immunity (Antibody determination)

| System | Component | Method | Kit/Manufacturer | Unit | Cut-off <sup>†</sup> | Laboratory* |
|---|---|---|---|---|---|---|
| Serum | Corynebacterium<br>diphtheriae.Diphtheria<br>Toxoid Ab.lgG | ELI | NA | IU/ml | 0.057 | GSK Biologicals<br>or designated<br>laboratory |
| Serum | Corynebacterium<br>diphtheriae.Diphtheria<br>Toxoid Ab | NEU<br>assay on<br>Vero<br>cells** | NA | IU/ml | 0.004 | GSK Biologicals<br>or designated<br>laboratory |
| Serum | Clostridium<br>tetani.Tetanus Toxoid<br>Ab.IgG | ELI | NA | IU/ml | 0.043 | GSK Biologicals or designated laboratory |
| Serum | Bordetella<br>pertussis.Pertussis<br>Toxin Ab.IgG | ELI | NA | IU/ml | 2.693 | GSK Biologicals or designated laboratory |
| Serum | Bordetella<br>pertussis.Filamentous<br>Hemaglutinin Ab.IgG | ELI | NA | IU/ml | 2.046 | GSK Biologicals<br>or designated<br>laboratory |
| Serum | Bordetella<br>pertussis.Pertactin<br>Ab.IgG | ELI | NA | IU/ml | 2.187 | GSK Biologicals<br>or designated<br>laboratory |

ELI: ELISA

**NEU: Neutralisation assay** 

NA: Not Applicable

IU/ml: International Units per millilitre

# 6.4. Analysis of safety

## 6.4.1. Analysis of safety planned in the protocol

The analysis will be based on the TVC.

- The percentage of subjects reporting each individual solicited local and general symptom during the 4-day (Day 1-4) follow-up period after booster vaccination will be tabulated. The same calculations will be done for each individual solicited symptom rated as grade 3 in intensity and for each individual solicited symptom assessed as causally related to vaccination.
- Occurrence of fever during the 4-day follow-up period after vaccination will be reported per 0.5°C cumulative increments.
  - In addition, the above analysis will also be done for sub groups based on age stratification (Refer Table 4) as an exploratory analysis.
- The percentage of subjects with at least one local symptom (solicited or unsolicited), with at least one general symptom (solicited or unsolicited) and with any symptom (solicited or unsolicited) during the 4-day (Day 1-4) follow-up period after booster

<sup>&</sup>lt;sup>†</sup>Assays for diphtheria, tetanus and pertussis were re-developed and re-validated as per most recent CBER recommendations (Guidance for Industry "Bioanalytical Method Validation" from September 2013). The new assay cutoff's that apply are listed in the table.

<sup>\*</sup>GSK Biologicals laboratory refers to the Clinical Laboratory Sciences (CLS) in Rixensart, Belgium and Wavre, Belgium.

<sup>\*\*</sup>Test on Vero-cells will be performed on pre- and post-vaccination samples with concentrations <0.1 IU/ml by ELISA.

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

vaccination will be tabulated with exact 95% CI after booster vaccination. The same calculations will be done for symptoms (solicited or unsolicited) rated as grade 3 in intensity, for symptoms (solicited or unsolicited) leading to medical consultation and for symptoms (solicited or unsolicited) assessed as causally related to vaccination.

- The percentage of subjects who started to receive at least one concomitant medication (i.e. any medication, antipyretic medication, prophylactic antipyretics) during the 4-day (Day 1-4) and 31-day (Day 1-31) follow-up period after vaccination will be tabulated with exact 95% CI.
- The verbatim reports of unsolicited AEs will be reviewed by a clinical research and development lead and the signs and symptoms will be coded according to MedDRA. Every verbatim term will be matched with the appropriate Preferred Term. The percentage of subjects with unsolicited AEs occurring within the 31-day (Day 1-31) follow-up period after booster dose with its exact 95% CI will be tabulated by Preferred Term. Similar tabulation will be done for unsolicited AEs rated as grade 3 and for unsolicited AEs with causal relationship to vaccination.
- Any large injection site reaction (for subjects <6 years of age defined as a swelling with a diameter of >50 mm and for subjects ≥6 years of age swelling with a diameter of >100 mm, noticeable diffuse swelling or noticeable increase in limb circumference) onset during the 4-day (Day 1-4) follow-up period after vaccination will be described in detail
- SAEs and withdrawal due to AEs and SAEs will be described in detail.

#### Handling of missing data:

- For a given subject and the analysis of solicited symptoms four days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore the analysis of the solicited symptoms based on the TVC will include only vaccinated subjects and doses with documented safety data (i.e., symptom screen completed).
- For analysis of unsolicited AEs, such as SAEs or AEs by primary Medical Dictionary for Regulatory Activities (MedDRA) term, and for the analysis of concomitant medications, all vaccinated subjects will be considered. Subjects, who do not report the event or the concomitant medication, will be considered as subjects without the event or the concomitant medication, respectively.
- For summaries reporting both solicited symptoms and unsolicited AEs, all vaccinated subjects will be considered. Subjects, who do not report the event or the concomitant medication, will be considered as subjects without the event or the concomitant medication, respectively.

#### 6.4.2. Additional considerations

The summary of each solicited symptoms and unsolicited adverse event will also be done for medically attended symptom/adverse event and for grade 3 causally related AE.

### 7. ANALYSIS INTERPRETATION

All analyses will be conducted in a descriptive manner.

#### 8. CONDUCT OF ANALYSES

Any deviation(s) or change(s) from the original statistical plan outlined in this protocol will be described and justified in the final study report.

## 8.1. Sequence of analyses

Analysis of the single booster dose will be performed at the end of the study when all data are available. An integrated clinical study report containing all data will be written and made available to the investigators.

## 8.2. Statistical considerations for interim analyses

All analyses will be conducted on final data and therefore no statistical adjustment for interim analyses is required.

| Description | Analysis<br>ID | Disclosure Purpose (IN=internal, CTRS=public posting, SR=study report and public posting) | Dry run<br>review<br>needed (Y/N) | Study Headline Summary (SHS)requiring expedited communication to upper management (Yes/No) | Reference for TFL |
|---|---|---|---|---|---|
| Final | E1_01 | SR | Yes | Yes | TFL TOC |

## 8.3. Statistical considerations for interim analyses

Not applicable

### 9. CHANGES FROM PLANNED ANALYSES

Not applicable

# 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The TFL TOC provides the list of tables/listings and figures needed for the study report. It also identifies the tables eligible for each analysis and their role (synopsis, in-text, post-text, SHS, CTRS,...). Note that all TFL aimed to be included as post-text are noted as post-text even if these are tabulation of individual data such as listing of SAE. The post-text material contains all source material for the study report and accordingly a post-text table may be redundant with an in-text table.

The mock tables referred under column named 'layout' can be found in Annex 3 of this SAP.

The following group name will be used in the TFLs, to be in line with the T-domains:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | dTpa Group | Boostrix |

# 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS

#### 11.1. Statistical Method References

The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413].

If some samples with anti-D concentrations < 0.1 IU/mL cannot be retested by VERO, VERO will be treated as left censored at 0.1 IU/mL and the Greenwoood formula for censored data will be used to estimate the percentage of subjects with anti-D antibody concentrations  $\geq$ 0.1 IU/mL by ELISA or anti-D concentrations  $\geq$ 0.01 IU/mL by VERO and its associated CI.

The 95% CI for GMTs/GMCs will be obtained within each group separately. The 95% CI for the mean of log-transformed titre/concentration will be first obtained assuming that log-transformed values were normally distributed with unknown variance. The 95% CI for the GMTs/GMCs will then be obtained by exponential-transformation of the 95% CI for the mean of log-transformed titre/concentration.

#### 11.2. Standard data derivation

#### 11.2.1. Date derivation

- SAS date derived from a character date: in case day is missing, 15 is used. In case day & month are missing, 30June is used.
- Onset day for an event (AE, medication, vaccination, ...): the onset day is the number of days between the last study vaccination & the onset/start date of the event. This is 0 for an event starting on the same day as a vaccination. See SAS date derived in case the start date of the event is incomplete.

## 11.2.2. Demography

Age: Age at the reference activity, computed as the number of complete weeks between the date of birth and the reference activity.

Conversion of weight to kg: the following conversion rule is used:

Weight in Kilogram= weight in Pounds / 2.2 + weight in ounces / 35.2

The result is rounded to 2 decimals.

Conversion of height to cm: the following conversion rule is used:

Height in Centimetres = Height in Feet \* 30.48+

Height in Inch \* 2.54

The result is rounded to the unit (ie no decimal).

Conversion of temperature to °C: the following conversion rule is used:

Temperature in °Celsius = ((Temperature in °Fahrenheit -32) \*5)/9

The result is rounded to 1 decimal.

## 11.2.3. Immunogenicity

- The geometric mean titres (GMTs)/geometric mean concentrations (GMCs) calculations will be performed by taking the anti-log of the mean of the log10 titre/concentration transformations. Antibody titres/concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off for the purpose of GMT/GMC calculation.
- In general, the assay cut-off is the value under which there is no quantifiable result available. For an assay with a specific 'assay cut\_off', numerical immuno result is derived from a character field (rawres):
  - If rawres is 'NEG' or '-' or '(-)', numeric result= assay cut off/2,
  - if rawres is 'POS' or '+' or '(+)', numeric result = assay cut off,

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

- if rawres is '< value' and value<=assay cut off, numeric result =assay cut off/2,</li>
- if rawres is '< value' and value>assay cut off, numeric result =value,
- if rawres is '> value' and value<assay cut off, numeric result =assay cut off/2,
- if rawres is '> value' and value>=assay cut off, numeric result =value,
- if rawres is '<= value' or '>= value' and value<assay cut\_off, numeric result</li>
   =assay cut\_off/2,
- if rawres is '<= value' or '>= value' and value>=assay cut\_off, numeric result =value,
- if rawres is a value < assay cut off, numeric result = assay cut off/2,</li>
- if rawres is a value >= assay cut off, numeric result = rawres,
- else numeric result is left blank.

## 11.2.4. Safety

For analysis of solicited, unsolicited adverse events (such as serious adverse events or adverse events by primary MedDRA term) and for the analysis of concomitant medications, all vaccinated subjects will be considered. Subjects who did not report the event or the concomitant medication will be considered as subjects without the event or the concomitant medication respectively.

The following rules will be used for the analysis of solicited symptoms:

- Subjects who documented the absence of a solicited symptom will be considered not having that symptom.
- Subjects who documented the presence of a solicited symptom and fully or
  partially recorded daily measurement over the solicited period will be included
  in the summaries at that dose and classified according to their maximum
  observed daily recording over the solicited period.
- Subjects who documented the presence of a solicited symptom without having recorded any daily measurement will be considered as having that symptom (at the lowest intensity).
- Intensity of the following solicited AEs will be assessed as described in Table 6 and below

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

Table 6 Intensity scales to be used by the parent(s)/LAR(s) for solicited symptoms during the solicited follow-up period

| Toddler/Child (<6 years) | | |
|---|---|---|
| Adverse Event | Intensity grade | Parameter |
| Pain at injection site | 0 | None |
| | 1 | Mild: Minor reaction to touch |
| | 2 | Moderate: Cries/protests on touch |
| | 3 | Severe: Cries when limb is moved/spontaneously painful |
| Redness at injection site | | Record greatest surface diameter in mm |
| Swelling at injection site | | Record greatest surface diameter in mm |
| Fever* | | Record temperature in °C |
| Irritability/Fussiness 0 | | Behaviour as usual |
| | 1 | Mild: Crying more than usual/no effect on normal activity |
| | 2 | Moderate: Crying more than usual/interferes with normal activit |
| | 3 | Severe: Crying that cannot be comforted/prevents normal |
| | | activity |
| Drowsiness | 0 | Behaviour as usual |
| | 1 | Mild: Drowsiness easily tolerated |
| | 2 | Moderate: Drowsiness that interferes with normal activity |
| | 3 | Severe: Drowsiness that prevents normal activity |
| Loss of appetite | 0 | Appetite as usual |
| | 1 | Mild: Eating less than usual/no effect on normal activity |
| | 2 | Moderate: Eating less than usual/interferes with normal activity |
| | 3 | Severe: Not eating at all |

<sup>\*</sup> Fever is defined as temperature ≥ 38.0°C. The preferred location for measuring temperature in this study will be the axilla

Table 7 Intensity scales for solicited symptoms in adults and children of six years of age or more

| Adult/Child (≥6 years) | | |
|---|---|---|
| Adverse Event | Intensity grade | Parameter |
| Pain at injection site | 0 | None |
| | 1 | Mild: Any pain neither interfering with nor preventing normal every day activities. |
| | 2 | Moderate: Painful when limb is moved and interferes with every day activities. |
| | 3 | Severe: Significant pain at rest. Prevents normal every day activities. |
| Redness at injection site | | Record greatest surface diameter in mm |
| Swelling at injection site | | Record greatest surface diameter in mm |
| Fever* | | Record temperature in °C |
| Headache | 0 | Normal |
| | 1 | Mild: Headache that is easily tolerated |
| | 2 | Moderate: Headache that interferes with normal activity |
| | 3 | Severe: Headache that prevents normal activity |
| Fatigue | 0 | Normal |
| | 1 | Mild: Fatigue that is easily tolerated |
| | 2 | Moderate: Fatigue that interferes with normal activity |
| | 3 | Severe: Fatigue that prevents normal activity |
| Gastrointestinal symptoms | 0 | Normal |
| (nausea, vomiting, diarrhoea and/or abdominal pain) | 1 | Mild: Gastrointestinal symptoms that are easily tolerated |
| | 2 | Moderate: Gastrointestinal symptoms that interfere with normal activity |
| | 3 | Severe: Gastrointestinal symptoms that prevent normal activity |

<sup>\*</sup> Fever is defined as temperature  $\geq$  38.0°C. The preferred location for measuring temperature in this study will be the axilla.

The maximum intensity of local injection site redness/swelling for toddlers and children <6 years of age will be scored at GSK Biologicals as follows:

| 0 | Absent |
|---|------------------|
| 1 | ≤5 mm |
| 2 | >5 mm and ≤20 mm |
| 3 | >20 mm |

The maximum intensity of local injection site redness/swelling for adults and children ≥6 years of age will be scored at GSK Biologicals as follows:

| ( | ) | Absent |
|----|---|-------------------|
| 1 | 1 | ≤20 mm |
| 2 | 2 | >20 mm and ≤50 mm |
| [3 | 3 | >50 mm |

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

The maximum intensity of fever will be scored at GSK Biologicals as follows:

| 0 | <38℃ |
|---|----------------------|
| 1 | ≥38.0 °C to ≤39.0 °C |
| 2 | >39.0 °C to ≤40.0 °C |
| 3 | >40.0℃ |

Note that for all tables described in this section, the way the percentage of subjects will be derived will depend on the event analysed (see table below for details). As a result, the N value will differ from one table to another.

| Event | N used for deriving % per subject for<br>Vaccination phase | N used for deriving % per dose for<br>Vaccination phase |
|---|---|---|
| Concomitant vaccination | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Solicited general symptom | All subjects with solicited symptoms documented as present or absent for at least one dose. | All doses with solicited symptoms documented as present or absent within 0-3 days post dose |
| Unsolicited symptom | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Concomitant medication | All subjects with study vaccine administered | All study visits with study vaccine administered |

For summaries by MedDRA primary preferred term combining solicited and unsolicited adverse events, solicited adverse events will be coded as per the following MedDRA codes

| Solicited symptom | Lower level term code | Corresponding<br>Lower level term<br>decode |
|---|---|---|
| Headache | 10019211 | Drowsiness |
| Fatigue | 10016256 | Fatigue |
| Gastrointestinal | 10017944 | |
| symptoms | | |
| Drowsiness | 10013649 | Drowsiness |
| Fever | 10016558 | Fever |
| Irritability/Fussiness | 10022998 | Irritability |
| Loss of appetite | 10003028 | Appetite lost |
| Pain at injection site | 10022086 | Injection site pain |
| Redness at injection | | Redness at |
| site | 10022098 | injection site |
| Swelling at | | Swelling at |
| injection site | 10053425 | injection site |

## 12. ANNEX 2: SUMMARY ON ELIMINATION CODES

Refer to section 5.2

### 13. ANNEX 3: STUDY SPECIFIC MOCK TFL

The following draft study specific mock TFLs will be used.

The data display, title and footnote are for illustration purpose and will be adapted to the study specificity such as one group and one dose for the study.

These templates were copied from recent studies. Note that there may be few changes between the study specific SAP mock TFL and the final TFLs. These editorial/minor changes will not lead to a SAP amendment.

Template 1 Number of subjects enrolled by center (Total Vaccinated Cohort)

| | Combo group | Control group | | Total |
|--------|-------------|---------------|-----|-------|
| Center | n | N | n | % |
| PPD | 20 | 21 | 41 | 9.1 |
| PPD | 27 | 28 | 55 | 12.2 |
| PPD | 7 | 7 | 14 | 3.1 |
| PPD | 16 | 16 | 32 | 7.1 |
| PPD | 27 | 26 | 53 | 11.8 |
| PPD | 26 | 26 | 52 | 11.5 |
| PPD | 25 | 25 | 50 | 11.1 |
| PPD | 23 | 24 | 47 | 10.4 |
| PPD | 22 | 22 | 44 | 9.8 |
| PPD | 24 | 25 | 49 | 10.9 |
| PPD | 7 | 7 | 14 | 3.1 |
| All | 224 | 227 | 451 | 100 |

<group description >

n = number of subjects included in each group or in total for a given center or for all centers

All = sum of all subjects in each group or in total (sum of all groups)

 $% = n/AII \times 100$ 

Template 2 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal at Visit 3 (Total Vaccinated Cohort)

| | HRV Liq | HRV<br>LYO | Total |
|---|---|---|---|
| Number of subjects vaccinated | 300 | 300 | 1200 |
| Number of subjects completed | 298 | 297 | 1193 |
| Number of subjects withdrawn | 2 | 3 | 7 |
| Reasons for withdrawal : | | | |
| Serious Adverse Event | 0 | 1 | 1 |
| Non-serious adverse event | 0 | 0 | 0 |
| Protocol violation | 0 | 0 | 0 |
| Consent withdrawal (not due to an adverse event) | 1 | 2 | 4 |
| Migrated/moved from study area | 1 | 0 | 2 |
| Lost to follow-up (subjects with incomplete vaccination course) | 0 | 0 | 0 |
| Lost to follow-up (subjects with complete vaccination course) | 0 | 0 | 0 |
| Others | 0 | 0 | 0 |

HRV LIQ = HRV vaccine liquid formulation

HRV LYO = HRV vaccine HRV Lyophilised formulation

Vaccinated = number of subjects who were vaccinated in the study

Completed = number of subjects who completed study visit 3

Withdrawn = number of subjects who did not come for study visit 3

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

Template 3 Number of subjects at each visit and list of withdrawn subjects (Total Vaccinated Cohort)

| Group | VISIT | N | Withdrawn<br>Subject numbers | Reason for withdrawal |
|---|---|---|---|---|
| HRV Liq | VISIT 1 | 508 | | |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. Pro | CONSENT WITHDRAWAL |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 2 | 504 | | |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | SERIOUS ADVERSE EXPERIENCE |
| | VISIT 3 | 501 | | |
| | | | no. P | MIGRATION FROM STUDY AREA |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. Pr | MIGRATION FROM STUDY AREA |
| | | | no. Pr | CONSENT WITHDRAWAL |
| | | | no. Pr | MIGRATION FROM STUDY AREA |
| | | | no. Pr | MIGRATION FROM STUDY AREA |
| | | | no. Pro | CONSENT WITHDRAWAL |
| | | | no. PPD | MIGRATION FROM STUDY AREA |
| | | | no. PPD | MIGRATION FROM STUDY AREA |
| | VISIT 4 | 492 | | |
| HRV Lyo | VISIT 1 | 257 | | |
| - | | | no. PP | PROTOCOL VIOLATION |
| | | | no. Pru | CONSENT WITHDRAWAL |
| | VISIT 2 | 255 | | |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 3 | 254 | | |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. Pr | LOST TO FOLLOW-UP |
| | | | no. Pr | LOST TO FOLLOW-UP |
| | | | no. Pr | CONSENT WITHDRAWAL |
| | | | no. Pr | MIGRATION FROM STUDY AREA |
| | | | no. Pro | LOST TO FOLLOW-UP |
| | | | no. PPD | ADVERSE EXPERIENCE |
| | VISIT 4 | 247 | | |

Template 4 Number of subjects enrolled into the study as well as the number of subjects excluded from ATP analyses with reasons for exclusion

| | | То | tal | | Н | RV L | IQ | HRV LYO | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Title | N n s | | | % | N n s | | | N n s | | s |
| Total enrolled cohort | 1200 | | | | 300 | | | 300 | | |
| TVC | 1200 | | | 100 | 300 | | | 300 | | |
| Administration of vaccine(s) | | 2 | 2 | | | 0 | 0 | | 0 | 0 |
| forbidden in the protocol | | | | | | | | | | |
| (code 1040) | | | | | | | | | | |
| Study vaccine dose not | | 73 | 73 | | | 23 | 23 | | 16 | 16 |
| administered according to | | | | | | | | | | |
| protocol (code 1070) | | | | | | | | | | |
| Initially seropositive or unknown | | 10 | 11 | | | 3 | 3 | | 1 | 1 |
| anti-rotavirus IgA antibody on | | | | | | | | | | |
| day of dose 1 (code 1500) | | | | | | | | | | |
| Protocol violation | | 1 | 1 | | | 1 | 1 | | 0 | 0 |
| (inclusion/exclusion criteria) | | | | | | | | | | |
| (code 2010) | | | | | | | | | | |
| Administration of any | | 1 | 1 | | | 0 | 0 | | 1 | 1 |
| medication forbidden by the | | | | | | | | | | |
| protocol (code 2040) | | | | | | | | | | |
| Underlying medical condition | | 1 | 1 | | | 0 | 0 | | 0 | 0 |
| forbidden by the protocol | | | | | | | | | | |
| (code 2050) | | | | | | | | | | |
| Concomitant infection not | | 0 | 1 | | | 0 | 0 | | 0 | 1 |
| related to the vaccine which | | | | | | | | | | |
| may influence immune | | | | | | | | | | |
| response (code 2070) | | | | | | | | | | |
| Non compliance with | | 14 | 16 | | | 6 | 7 | | 3 | 4 |
| vaccination schedule (including | | | | | | | | | | |
| wrong and unknown dates) | | | | | | | | | | |
| (code 2080) | | | | | | | | | | |
| Non compliance with blood | | 12 | 16 | | | 3 | 5 | | 4 | 5 |
| sampling schedule (including | | | | | | | | | | |
| wrong and unknown dates) | | | | | | | | | | |
| (code 2090) | | | | | | | | | | |
| Essential serological data | | 87 | 95 | | | 20 | 22 | | 23 | 26 |
| missing (code 2100) | | | | | | | | | | |
| Subjects with incomplete study | | 1 | 1 | | | 0 | 0 | | 0 | 0 |
| vaccination schedule but with | | | | | | | | | | |
| post serological result (code | | | | | | | | | | |
| 2500) | | | | | | | | | | |
| ATP | 998 | | | 83.2 | 244 | | | 252 | | |

HRV LIQ = HRV vaccine liquid formulation Lot C HRV LYO = HRV vaccine HRV Lyophilised formulation Note: Subjects may have more than one elimination code assigned

n = number of subjects with the elimination code assigned excluding subjects who have been assigned a lower elimination code number

s = number of subjects with the elimination code assigned

<sup>% =</sup> percentage of subjects in the per protocol set (ATP) relative to the TVC (ES)

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

Template 5 Deviations from specifications for age and intervals between study visits (Total Vaccinated Cohort)

| | | Age | VA | AC_1-SER_2 |
|---|---|---|---|---|
| Group | | Protocol | Protocol | Adapted |
| - | | from 10 to 15 year | from 30 to 48 days | from 21 to 48 days |
| dTpaNew Group | N | 335 | 329 | 329 |
| | n | 0 | 11 | 8 |
| | % | 0.0 | 3.3 | 2.4 |
| | range | 10 to 15 | 28 to 74 | 28 to 74 |
| dTpaPre Group | N | 336 | 329 | 329 |
| | n | 0 | 10 | 8 |
| | % | 0.0 | 3.0 | 2.4 |
| | range | 10 to 15 | 29 to 95 | 29 to 95 |

HRV LIQ = HRV vaccine liquid formulation Lot A

HRV LIQ = HRV vaccine liquid formulation Lot B

HRV LIQ = HRV vaccine liquid formulation Lot C

HRV LYO = HRV vaccine HRV Lyophilised formulation

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

Adapted = interval used for defining the ATP cohorts for immunogenicity

N = total number of subjects with available results

n(%) = number(percentage) of subjects with results outside of the interval

range = minimum-maximum for age and intervals

VAC = vaccination

SER = Blood Sampling

Template 6 Summary of demographic characteristics (ATP cohort for Immunogenicity)

| | | dTpaNe<br>Group<br>N = 33 | ) | dTpaPre<br>Group<br>N = 336 | | Tota<br>N = 67 | - |
|---|---|---|---|---|---|---|---|
| Characteristics | Parameters or Categories | Value or n | % | Value or<br>n | % | Value or n | % |
| Age (years) at vaccination dose: 1 | Mean | 11.9 | - | 11.9 | - | 11.9 | - |
| | SD | 1.59 | - | 1.61 | - | 1.60 | - |
| | Median | 12.0 | - | 12.0 | - | 12.0 | - |
| | Minimum | 10 | - | 10 | - | 10 | - |
| | Maximum | 15 | - | 15 | - | 15 | - |
| Gender | Female | 179 | 53.4 | 178 | 53.0 | 357 | 53.2 |
| | Male | 156 | 46.6 | 158 | 47.0 | 314 | 46.8 |
| Geographic Ancestry | African Heritage / African American | 1 | 0.3 | 1 | 0.3 | 2 | 0.3 |
| | American Indian or Alaskan Native | 146 | 43.6 | 149 | 44.3 | 295 | 44.0 |
| | White - Arabic / North African | 1 | 0.3 | 0 | 0.0 | 1 | 0.1 |
| | Heritage | | | | | | |
| | White - Caucasian / European<br>Heritage | 9 | 2.7 | 12 | 3.6 | 21 | 3.1 |
| | Other (Hispanic) | 178 | 53.1 | 174 | 51.8 | 352 | 52.5 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

N = total number of subjects

n(%) = Number(percentage) of subjects in a given category

Value = value of the considered parameter

SD = standard deviation

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

**Template 7** Summary of vital signs characteristics (Total Vaccinated Cohort)

| | | dTpaNew Group<br>(N = 335) | dTpaPre Group<br>(N = 336) | Total<br>(N = 671) |
|---|---|---|---|---|
| Characteristics | Parameters | Value | Value | Value |
| Height (km) | Mean | 152.6 | 151.5 | 152.1 |
| | SD | 10.48 | 10.44 | 10.47 |
| | Median | 152.0 | 151.5 | 152.0 |
| | Minimum | 112.0 | 126.0 | 112.0 |
| | Maximum | 189.0 | 187.0 | 189.0 |
| | Unknown | 0 | 0 | 0 |
| Weight (kg) | Mean | 49.7 | 48.8 | 49.2 |
| | SD | 13.23 | 13.61 | 13.42 |
| | Median | 47.0 | 47.1 | 47.0 |
| | Minimum | 28.0 | 19.4 | 19.4 |
| | Maximum | 99.0 | 110.0 | 110.0 |
| | Unknown | 0 | 0 | 0 |
| BMI (kg/m²) | Mean | 21.1 | 20.9 | 21.0 |
| | SD | 3.92 | 3.91 | 3.92 |
| | Median | 20.6 | 20.4 | 20.4 |
| | Minimum | 11.9 | 9.8 | 9.8 |
| | Maximum | 33.5 | 34.0 | 34.0 |
| | Unknown | 0 | 0 | 0 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

N = total number of subjects

Value = value of the considered parameter

SD = standard deviation

Height (cm) = Height expressed in centimeters

Weight (kg) = Weight expressed in kilograms

BMI (kg/m²) = Body Mass Index expressed in kilograms per meter square

#### **Template 8 Study population (Total Vaccinated Cohort)**

| Number of subjects | Combo<br>group | Control group |
|---|---|---|
| Planned, N | 225 | 225 |
| Randomised, N (Total Vaccinated Cohort) | 224 | 227 |
| Completed, n (%) | 224 (100) | 227 (100) |
| Demographics | Combo | Control |
| | group | group |
| N (Total Vaccinated Cohort) | 224 | 227 |
| Females :Males | 97:127 | 115:112 |
| Mean Age, weeks (SD) | 8.8 (1.1) | 8.8 (1.1) |
| Median Age, weeks (minimum, maximum) | 9 (7, 11) | 9 (7, 11) |
| Most frequent race: Asian - East Asian Heritage, n (%) | 224 (100) | 226 (99.6) |

Combo group = Subjects received DTPa-IPV/Hib vaccine as a single injection at 2, 4 and 6 months of age

Control group = Subjects received DTPa-IPV and Hib vaccines at different injection sites at 2, 4 and 6 months of age

N = Total number of subjects enrolled in the study

n/% = Number/percentage of subjects in a given category

SD = Standard Deviation

MeaAge = Age calculated from Date of birth to first study vaccination

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

Template 9 Seropositivity and seroprotection rates and GMCs for anti-diphtheria and anti-tetanus antibodies before and one month after the booster vaccination (ATP cohort for immunogenicity)

| | | | | ≥ | assay | / cut- | off* | | ≥ 0.1 | IU/ml | | | GMC | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95% | 6 CI | | | 95% | 6 CI | | 959 | % CI |
| Antibody | Group | Timing | N | n | % | LL | UL | n | % | LL | UL | value | LL | UL |
| anti-diphtheria | dTpaNew Group | PRE | 321 | 284 | 88.5 | 84.5 | 91.8 | 83 | 25.9 | 21.2 | 31.0 | 0.472 | 0.403 | 0.553 |
| | | POST | 321 | 320 | 99.7 | 98.3 | 100 | 315 | 98.1 | 96.0 | 99.3 | 6.784 | 6.178 | 7.450 |
| | dTpaPre Group | PRE | 319 | 286 | 89.7 | 85.8 | 92.8 | 89 | 27.9 | 23.0 | 33.2 | 0.456 | 0.392 | 0.530 |
| | | POST | 319 | 319 | 100 | 98.9 | 100 | 310 | 97.2 | 94.7 | 98.7 | 6.493 | 5.915 | 7.128 |
| anti-tetanus | dTpaNew Group | PRE | 321 | 311 | 96.9 | 94.3 | 98.5 | 151 | 47.0 | 41.5 | 52.7 | 0.956 | 0.835 | 1.095 |
| | | POST | 321 | 321 | 100 | 98.9 | 100 | 321 | 100 | 98.9 | 100 | 18.937 | 17.313 | 20.713 |
| | dTpaPre Group | PRE | 319 | 314 | 98.4 | 96.4 | 99.5 | 143 | 44.8 | 39.3 | 50.5 | 0.899 | 0.789 | 1.026 |
| ı | | POST | 319 | 319 | 100 | 98.9 | 100 | 319 | 100 | 98.9 | 100 | 18.515 | 16.851 | 20.342 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

Seroprotection=anti-diphtheria and anti-tetanus antibody concentration ≥0.1 IU/mL

\*Assay cut-off is 0.057 IU/mL and 0.043 IU/mL for anti-diphtheria and anti-tetanus respectively

GMC = geometric mean antibody concentration calculated on all subjects

N = number of subjects with available results

n(%)=number(percentage) of subjects with antibody concentrations above the specified cut-off

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

PRE=Pre-booster blood sampling time point

POST=Post-booster blood sampling time point

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

Template 10 Booster responses for anti-PT, anti-FHA and anti-PRN antibody concentration one month after the booster vaccination (ATP cohort for immunogenicity)

| | | | | | Booste | r respor | ıse |
|---|---|---|---|---|---|---|---|
| | | | | | | | 5% CI |
| Antibody | Group | Pre-vaccination status | n | % | LL | UL | |
| anti-PT | dTpaNew Group | S- | 142 | 135 | 95.1 | 90.1 | 98.0 |
| | | S+ (< 4*assay cut-off) | 104 | 103 | 99.0 | 94.8 | 100 |
| | | S+ (≥4*assay cut-off) | 71 | 60 | 84.5 | 74.0 | 92.0 |
| | | Total | 317 | 298 | 94.0 | 90.8 | 96.4 |
| | dTpaPre Group | S- | 143 | 131 | 91.6 | 85.8 | 95.6 |
| | | S+ (<4*assay cut-off) | 114 | 112 | 98.2 | 93.8 | 99.8 |
| | | S+ (≥4*assay cut-off) | 61 | 52 | 85.2 | 73.8 | 93.0 |
| | | Total | 318 | 295 | 92.8 | 89.3 | 95.4 |
| anti-FHA | dTpaNew Group | S- | 6 | 6 | 100 | 54.1 | 100 |
| | | S+ (<4*assay cut-off) | 57 | 57 | 100 | 93.7 | 100 |
| | | S+ (≥4*assay cut-off) | 251 | 242 | 96.4 | 93.3 | 98.3 |
| | | Total | 314 | 305 | 97.1 | 94.6 | 98.7 |
| | dTpaPre Group | S- | 5 | 5 | 100 | 47.8 | 100 |
| | | S+ (<4*assay cut-off) | 55 | 55 | 100 | 93.5 | 100 |
| | | S+ (≥4*assay cut-off) | 255 | 244 | 95.7 | 92.4 | 97.8 |
| | | Total | 315 | 304 | 96.5 | 93.8 | 98.2 |
| anti-PRN | dTpaNew Group | S- | 52 | 50 | 96.2 | 86.8 | 99.5 |
| | | S+ (<4*assay cut-off) | 152 | 151 | 99.3 | 96.4 | 100 |
| | | S+ (≥4*assay cut-off) | 117 | 114 | 97.4 | 92.7 | 99.5 |
| | | Total | 321 | 315 | 98.1 | 96.0 | 99.3 |
| | dTpaPre Group | S- | 47 | 47 | 100 | 92.5 | 100 |
| | | S+ (<4*assay cut-off) | 159 | 159 | 100 | 97.7 | 100 |
| | | S+ (≥4*assay cut-off) | 112 | 111 | 99.1 | 95.1 | 100 |
| | | Total | 318 | 317 | 99.7 | 98.3 | 100 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

Total = subjects either seropositive or seronegative at pre-vaccination

S- = seronegative subjects (antibody concentration below assay cut off for anti-PT, anti-FHA, anti-PRN)

S+ = seropositive (antibody concentration below assay cut off for anti-PT, anti-FHA, anti-PRN)

Booster response to PT, FHA and PRN antigens is defined as:

- initially seronegative subjects (pre-booster antibody concentration below the assay cut-off) with an increase
  of at least four times the assay cut-off one month after vaccination.
- initially seropositive subjects with anti-body concentration < four times the assay cut-off with an increase of at least four times the pre-booster antibody concentration one month after vaccination
- initially seropositive subjects with anti-body concentration ≥ four times the assay cut-off with an increase of at least two times the pre-booster antibody concentration one month after vaccination

Assay cut-off is 2.693 IU/mL, 2.046 IU/mL and 2.187 IU/mL for anti-PT, FHA and PRN respectively

N = number of subjects with both pre- and post-vaccination results available

n(%) = number(percentage) of subjects with a booster response

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

S- = Initially seronegative subjects prior to vaccination

S+ = Initially seropositive subjects prior to vaccination

Template 11 Reverse cumulative curve for anti-diphtheria antibody concentration one month after the booster vaccination (ATP cohort for immunogenicity)



dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

# Template 12 Seroprotection rate for anti-Diphtheria antibody concentration by ELISA and VERO NEUTRALISATION (ATP cohort)

| | | | conce<br>belov | LISA<br>Intrations<br>In the 0.1<br>IJ/ml | below the<br>subject<br>concentr | concentrations 0.01 IU/ml among cts with ELISA ations below the 0.1 IU/ml | Neutra conce<br>below the 0.<br>among subje<br>ELISA re | 01 IU/ml<br>ects with | prote | stimate<br>oportion<br>cted su<br>and its 9 | n of<br>bjects |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Group | Timing | N | n/N | % | n'/N' | % | n/N x n'/N' | % | SP | LL | UL |
| (each group) | Pre post | | | | | | | | | | |

Boostrix group= Subjects who had received GSK Biologicals' Tdap vaccine (Boostrix) in study 106316 and a second dose of Tdap vaccine (Boostrix) at Year 9 Visit 6

Adacel group= Subjects who had received Sanofi Pasteurs' Tdap vaccine (Adacel) in study 106316 and a second dose of Tdap vaccine (Boostrix) at Year 9 Visit 6

N = number of subjects tested by ELISA

N' = number of subjects with ELISA concentrations below the 0.1 IU/ml who were tested by Vero

% = proportion of subjects with concentrations below the considered cut-off (0.1 IU/ml for ELISA and 0.01 IU/ml for

VERO) n/N x n'/N' = the multiplication of the two proportions = overall seronegativity for anti-Diphtheria

Overall = based on both the ELISA and the Vero-cell neutralisation testing

95% CI = exact 95% confidence interval; LL = lower limit, UL = upper limit

Pre= blood sampling, at Month 0 before vaccination

post= blood sampling, one moth after vaccination

SP= proportion of subjects with either ELISA concentrations above 0.1 IU/ml or Neutra concentration above 0.01 IU/mL

Template 13 Compliance in returning symptom information (Total Vaccinated Cohort)

| Group | Number<br>of<br>doses | Doses NOT according to protocol | Number<br>of<br>general SS | Compliance<br>%<br>general SS | Number<br>of<br>local SS | Compliance<br>%<br>local SS |
|---|---|---|---|---|---|---|
| dTpaNew Group | 335 | 0 | 330 | 98.5 | 330 | 98.5 |
| dTpaPre Group | 336 | 1 | 329 | 97.9 | 329 | 97.9 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

SS = Symptom screens/sheets used for the collection of local and general solicited AEs

Compliance % = (number of doses with symptom screen/sheet return / number of administered doses) X 100
201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

Template 14 Incidence and nature of grade 3 symptoms (solicited and unsolicited) reported during the 4-day (Days 0-3) period after vaccination following each dose and overall (Total Vaccinated Cohort)

| | | Any symptom | | | | | Gene | ral syr | nptom | S | Local symptoms | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% | % CI | | | | 959 | % CI | | | | 959 | % CI |
| Group | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| dTpaNew Group | 335 | 264 | 78.8 | 74.0 | 83.1 | 335 | 134 | 40.0 | 34.7 | 45.5 | 335 | 250 | 74.6 | 69.6 | 79.2 |
| dTpaPre Group | 336 | 279 | 83.0 | 78.6 | 86.9 | 336 | 151 | 44.9 | 39.5 | 50.4 | 336 | 264 | 78.6 | 73.8 | 82.8 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Template 15 Incidence of solicited local symptoms reported during the 4-day (Days 0-3) period after vaccination following each dose and overall (Total Vaccinated Cohort)

| | | | dT | paNew | Group | | | dΤ | paPre | Group | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | • | 95 | % CI | | | | 95 | % CI |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL |
| Pain | All | 330 | 237 | 71.8 | 66.6 | 76.6 | 329 | 248 | 75.4 | 70.4 | 79.9 |
| | Grade 3 | 330 | 24 | 7.3 | 4.7 | 10.6 | 329 | 20 | 6.1 | 3.8 | 9.2 |
| | Medical advice | 330 | 0 | 0.0 | 0.0 | 1.1 | 329 | 0 | 0.0 | 0.0 | 1.1 |
| Redness (mm) | All | 330 | 113 | 34.2 | 29.1 | 39.6 | 329 | 94 | 28.6 | 23.8 | 33.8 |
| | Grade 3 | 330 | 4 | 1.2 | 0.3 | 3.1 | 329 | 1 | 0.3 | 0.0 | 1.7 |
| | Medical advice | 330 | 0 | 0.0 | 0.0 | 1.1 | 329 | 0 | 0.0 | 0.0 | 1.1 |
| Swelling (mm) | All | 330 | 98 | 29.7 | 24.8 | 34.9 | 329 | 90 | 27.4 | 22.6 | 32.5 |
| - ' ' | Grade 3 | 330 | 6 | 1.8 | 0.7 | 3.9 | 329 | 5 | 1.5 | 0.5 | 3.5 |
| | Medical advice | 330 | 0 | 0.0 | 0.0 | 1.1 | 329 | 0 | 0.0 | 0.0 | 1.1 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

N = number of subjects with the administered dose

n(%)= number(percentage) of subjects presenting at least one type of symptom whatever the study vaccine administered

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

N = number of subjects with the documented dose

n(%)= number(percentage) of subjects reporting the symptom at least once

<sup>95%</sup>CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

## Template 16 Incidence of solicited general symptoms reported during the 4-day (Days 0-3) post-vaccination period (Total Vaccinated Cohort)

| | | | dΤι | paNew | Grou | р | | dΤμ | aPre | Group | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 | % CI | | • | | 95 | % CI |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL |
| Fatigue | All | 330 | 83 | 25.2 | 20.6 | 30.2 | 329 | 86 | 26.1 | 21.5 | 31.2 |
| | Grade 3 | 330 | 7 | 2.1 | 0.9 | 4.3 | 329 | 4 | 1.2 | 0.3 | 3.1 |
| | Related | 330 | 77 | 23.3 | 18.9 | 28.3 | 329 | 83 | 25.2 | 20.6 | 30.3 |
| | Medical advice | 330 | 1 | 0.3 | 0.0 | 1.7 | 329 | 1 | 0.3 | 0.0 | 1.7 |
| Gastrointestinal | All | 330 | 32 | 9.7 | 6.7 | 13.4 | 329 | 42 | 12.8 | 9.4 | 16.9 |
| | Grade 3 | 330 | 3 | 0.9 | 0.2 | 2.6 | 329 | 3 | 0.9 | 0.2 | 2.6 |
| | Related | 330 | 29 | 8.8 | 6.0 | 12.4 | 329 | 40 | 12.2 | 8.8 | 16.2 |
| | Medical advice | 330 | 2 | 0.6 | 0.1 | 2.2 | 329 | 1 | 0.3 | 0.0 | 1.7 |
| Headache | All | 330 | 88 | 26.7 | 22.0 | 31.8 | 329 | 108 | 32.8 | 27.8 | 38.2 |
| | Grade 3 | 330 | 5 | 1.5 | 0.5 | 3.5 | 329 | 3 | 0.9 | 0.2 | 2.6 |
| | Related | 330 | 80 | 24.2 | 19.7 | 29.2 | 329 | 103 | 31.3 | 26.3 | 36.6 |
| | Medical advice | 330 | 2 | 0.6 | 0.1 | 2.2 | 329 | 1 | 0.3 | 0.0 | 1.7 |
| Temperature/(Axillary) (°C) | All | 330 | 9 | 2.7 | 1.3 | 5.1 | 329 | 6 | 1.8 | 0.7 | 3.9 |
| , , , , | ≥37.5 | 330 | 9 | 2.7 | 1.3 | 5.1 | 329 | 6 | 1.8 | 0.7 | 3.9 |
| | >38.0 | 330 | 5 | 1.5 | 0.5 | 3.5 | 329 | 1 | 0.3 | 0.0 | 1.7 |
| | >38.5 | 330 | 3 | 0.9 | 0.2 | 2.6 | 329 | 1 | 0.3 | 0.0 | 1.7 |
| | >39.0 | 330 | 2 | 0.6 | 0.1 | 2.2 | 329 | 0 | 0.0 | 0.0 | 1.1 |
| | Related | 330 | 7 | 2.1 | 0.9 | 4.3 | 329 | 6 | 1.8 | 0.7 | 3.9 |
| | Medical advice | 330 | 2 | 0.6 | 0.1 | 2.2 | 329 | 0 | 0.0 | 0.0 | 1.1 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

N = number of subjects with the documented dose

n(%)= number(percentage) of subjects reporting the symptom at least once

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

Related = Symptoms which is assessed by the investigator as related to vaccination

Grade3\*Related = Grade 3 symptom which is assessed by the investigator as related to vaccination

Grade 3 For Headache: Headache that prevented normal activity

For Fatigue: Fatigue that prevented normal activity

For Gastrointestinal symptoms: Gastrointestinal symptoms that prevented normal activity

For Fever: >39.0 °C

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

Template 17 Percentage of subjects with grade 3 unsolicited symptoms classified by MedDRA SOC and PT from Day 0 to Day 30 after any vaccination (Total Vaccinated Cohort)

| Primary System Organ | Preferred | | | LIQ<br>298 | | | | / LIQ<br>: 302 | | | | LIQ<br>300 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Class (CODE) | Term (CODE) | | | 95% | 6 CI | | | 95 | % CI | | | 95 | % CI |
| , , | , , | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| At least one symptom | | 24 | 8.1 | 5.2 | 11.7 | 26 | 8.6 | 5.7 | 12.4 | 33 | 11.0 | 7.7 | 15.1 |
| Ear and labyrinth | Ear pain | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| disorders (10013993) | (10014020) | | | | | | | | | | | | |
| Eye disorders (10015919) | Conjunctivitis (10010741) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 1 | 0.3 | 0.0 | 1.8 |
| Gastrointestinal disorders (10017947) | Diarrhoea (10012735) | 0 | 0.0 | 0.0 | 1.2 | 2 | 0.7 | 0.1 | 2.4 | 1 | 0.3 | 0.0 | 1.8 |
| disorders (10011341) | Flatulence<br>(10016766) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 2 | 0.7 | 0.1 | 2.4 |
| General disorders and administration site conditions (10018065) | Injection site erythema (10022061) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Injection site pain (10022086) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Injection site<br>swelling<br>(10053425) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Irritability<br>(10022998) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 1 | 0.3 | 0.0 | 1.8 |
| | Pyrexia (10037660) | 4 | 1.3 | 0.4 | 3.4 | 3 | 1.0 | 0.2 | 2.9 | 4 | 1.3 | 0.4 | 3.4 |
| Immune system disorders (10021428) | Hypersensitivit y (10020751) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| Infections and infestations (10021881) | Bronchitis<br>(10006451) | 2 | 0.7 | 0.1 | 2.4 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Ear infection<br>(10014011) | 1 | 0.3 | 0.0 | 1.9 | 3 | 1.0 | 0.2 | 2.9 | 2 | 0.7 | 0.1 | 2.4 |
| | Exanthema subitum (10015586) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| | Eye infection (10015929) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Gastroenteritis (10017888) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Impetigo<br>(10021531) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Influenza<br>(10022000) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| | Laryngitis<br>(10023874) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Otitis media (10033078) | 5 | 1.7 | 0.5 | 3.9 | 6 | 2.0 | 0.7 | 4.3 | 11 | 3.7 | 1.8 | 6.5 |
| | Perianal<br>abscess<br>(10034447) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

| | | | HRV | LIQ | | | HRV | / LIQ | | . , | | / LIQ | 11 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Primary System Organ | Preferred | | | 298 | | | | 302 | | | | 300 | |
| Class (CODE) | Term (CODE) | | | 95% | 6 CI | | | 95 | % CI | | | | % CI |
| , , | , , | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| | Pneumonia<br>(10035664) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| | Respiratory<br>tract infection<br>(10062352) | 3 | 1.0 | 0.2 | 2.9 | 2 | 0.7 | 0.1 | 2.4 | 0 | 0.0 | 0.0 | 1.2 |
| | Respiratory<br>tract infection<br>viral<br>(10062106) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Rhinitis<br>(10039083) | 2 | 0.7 | 0.1 | 2.4 | 1 | 0.3 | 0.0 | 1.8 | 3 | 1.0 | 0.2 | 2.9 |
| | Upper respiratory tract infection (10046306) | 2 | 0.7 | 0.1 | 2.4 | 5 | 1.7 | 0.5 | 3.8 | 7 | 2.3 | 0.9 | 4.7 |
| | Varicella<br>(10046980) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 2 | 0.7 | 0.1 | 2.4 |
| Psychiatric disorders (10037175) | Crying (10011469) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| Respiratory, thoracic and mediastinal disorders (10038738) | Cough<br>(10011224) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 6 | 2.0 | 0.7 | 4.3 |
| | Nasal<br>congestion<br>(10028735) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Rales<br>(10037833) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| Skin and subcutaneous tissue disorders (10040785) | Dermatitis<br>allergic<br>(10012434) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| | Eczema<br>(10014184) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Rash<br>(10037844) | 2 | 0.7 | 0.1 | 2.4 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |

HRV LIQ = HRV vaccine liquid formulation Lot A

HRV LIQ = HRV vaccine liquid formulation Lot B

HRV LIQ = HRV vaccine liquid formulation Lot C

N = number of subjects with at least one administered dose n/% = number/percentage of subjects reporting at least once a specified unsolicited symptom

At least one symptom = number of subjects reporting at least one unsolicited symptom, whatever the MedDRA PT

95% CI = exact 95% Confidence Interval, LL = Lower Limit, UL = Upper Limit

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

# Template 18 Number (%) of subjects with serious adverse events from first study vaccination up to Visit 3 including number of events reported (Total Vaccinated Cohort)

| | | | | Gr 1<br>N = | | | Gr2<br>N = | |
|---|---|---|---|---|---|---|---|---|
| Type of Event | Primary System Organ<br>Class | Preferred Term (CODE) | n* | n | % | n* | n | % |
| SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Related SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Fatal SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Related fatal SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |

Gr 1 = Group 1 description

Gr 2 = Group 2 description

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

## Template 19 Subjects with Serious Adverse Events reported up to Visit 2 (Total Vaccinated Cohort)

| Sub.<br>No. | Case Id | Age at onset (Week) | Sex | Verbatim | Preferred term | System Organ<br>Class | MA<br>type | Dose | Day of onset | Duration | Causality | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| P<br>P | PPD | | М | Kawasaki's<br>disease | Kawasaki's<br>disease | Infections and infestations | НО | 1 | 12 | 29 | N | Recovered/resolved |
| PP<br>D | PPD | 18 | M | Influenza-b | Influenza | Infections and infestations | НО | 2 | 2 | 5 | N | Recovered/resolved |
| PP<br>D | PPD | 17 | M | Acute gastroenteritis | Gastroenteritis | Infections and infestations | НО | 2 | 9 | 5 | N | Recovered/resolved |
| PP<br>D | PPD | 17 | F | Infantile spasms | Infantile spasms | Nervous system disorders | НО | 2 | 2 | 51 | N | Recovered/resolved with sequelae |
| PP<br>D | PPD | 21 | М | Rs-virus<br>bronchiolitis | Respiratory<br>syncytial virus<br>bronchiolitis | Infections and infestations | НО | 2 | 30 | 16 | N | Recovered/resolved |
| PP<br>D | PPD | 13 | М | Gastroenteritis | Gastroenteritis | Infections and infestations | НО | 1 | 25 | 6 | N | Recovered/resolved |
| PP<br>D | PPD | 22 | М | Pneumonia | Pneumonia | Infections and infestations | НО | 2 | 32 | 13 | N | Recovered/resolved |
| | | 23 | | Middle ear infection | Otitis media | Infections and infestations | НО | 2 | 37 | 8 | N | Recovered/resolved |
| PP<br>D | PPD | 14 | F | Secretory otitis media | Otitis media | Infections and infestations | НО | 1 | 7 | 25 | N | Recovered/resolved |
| PPD | PPD | 20 | M | Viral pneumonia | Pneumonia viral | Infections and infestations | НО | 2 | 13 | 23 | N | Recovered/resolved |
| PPD | PPD | 14 | М | Middle ear infection, left | Otitis media | Infections and infestations | НО | 1 | 19 | 8 | N | Recovered/resolved |
| | | 14 | | Pneumonia | Pneumonia | Infections and infestations | НО | 1 | 19 | 8 | N | Recovered/resolved |
| PPD | PPD | 13 | М | Acute lymphadenitis | Lymphadenitis | Blood and lymphatic system disorders | НО | 1 | 13 | 22 | N | Recovered/resolved |
| PPD | PPD | 10 | F | Pyelonephritis acute | Pyelonephritis acute | Infections and infestations | НО | 1 | 6 | 12 | N | Recovered/resolved |
| PPD | PPD | 19 | М | Laryngitis | Laryngitis | Infections and infestations | НО | 2 | 11 | 7 | N | Recovered/resolved |
| PPD | PPD | 14 | М | Bronchitis acuta | Bronchitis | Infections and | НО | 1 | 23 | 12 | N | Recovered/resolved |

## 201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

| Sub.<br>No. | Case Id | Age at onset (Week) | | Verbatim | Preferred term | System Organ<br>Class | MA<br>type | Dose | Day of onset | Duration | Causality | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | infestations | | | | | | |
| PPD | PPD | 19 | М | Bronchiolitis acuta | Bronchiolitis | Infections and infestations | НО | 2 | 26 | 7 | N | Recovered/resolved |
| PPD | PPD | 19 | F | Laryngitis acuta | Laryngitis | Infections and infestations | НО | 2 | 7 | 4 | N | Recovered/resolved |
| PPD | PPD | 18 | F | Laryngitis | Laryngitis | Infections and infestations | НО | 2 | 7 | 4 | N | Recovered/resolved |
| PPD | PPD | 14 | F | Gastroenteritis | Gastroenteritis | Infections and infestations | НО | 1 | 22 | 7 | N | Recovered/resolved |

MA = medical attention

HO = hospitalisation

Dose = dose given prior to the start of the SAE
Day of onset = number of days since last study vaccine dose

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

Template 20 Number and percentage of subjects who started at least one concomitant medication from Day 0 to Day 7 (Total Vaccinated Cohort)

| | | ď | TpaNew | Group | | | d | TpaPre | Group | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | _ | 9 | 5% CI | | | - | 9 | 5% CI |
| | N | n | % | LL | UL | N | n | % | LL | UL |
| Any | 335 | 41 | 12.2 | 8.9 | 16.2 | 336 | 43 | 12.8 | 9.4 | 16.8 |
| Any antipyretic | 335 | 37 | 11.0 | 7.9 | 14.9 | 336 | 41 | 12.2 | 8.9 | 16.2 |
| Prophylactic antipyretic | 335 | 2 | 0.6 | 0.1 | 2.1 | 336 | 2 | 0.6 | 0.1 | 2.1 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

Template 21 Solicited and Unsolicited symptoms experienced by subjects classified by MedDRA Primary System Organ Class and Preferred Term within the 31-day (Days 0-30) post-vaccination period - SAE excluded (Total vaccinated cohort)

| | | Н | IPV_<br>N : | _ | MMI | R_D<br>N = | |
|---|---|---|---|---|---|---|---|
| <b>Primary System Organ Class (CODE)</b> | Preferred Term (CODE | n* | n | % | n* | n | % |
| At least one symptom | | | | | | | |
| <each soc=""></each> | <each pt="" term=""></each> | | | | | | |

HPV\_2D = females aged 4-6 years who received two doses of HPV-16/18 L1 VLP AS04 vaccine at Day 0 and Month 6 MMR\_DTPa = females aged 4-6 years who received MMR vaccine at Day 0 and DTPa vaccine at Month 6 At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n/% = number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Template 22 Minimum and maximum activity dates (TVC)

| Visit | Minimum date | Maximum date |
|-------|--------------|--------------|
| 1 | 19JUN2007 | 29DEC2007 |
| 2 | 24JUL2007 | 08FEB2008 |
| 3 | 24AUG2007 | 18MAR2008 |
| 4 | 25MAR2008 | 22NOV2008 |
| 5 | 24MAR2009 | 31MAR2009* |

<sup>\*</sup>Database Lock Date = 31MAR2009

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

N = number of subjects with the administered dose

n(%)= number(percentage) of subjects who started to take the specified concomitant medication at least once during the mentioned period

<sup>95%</sup> CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

n\* = number of events reported

#### Template 23 Number of enrolled subjects by age category (TVC)

| | | Gr 1<br>N = | Gr 2<br>N = | Gr 3<br>N = | Total<br>N = |
|---|---|---|---|---|---|
| Characteristics | Categories | n | n | n | n |
| Age category | In utero | | | | |
| | Preterm newborn infants | | | | |
| | (gestational age < 37 wks) | | | | |
| | Newborns (0-27 days) | | | | |
| | Infants and toddlers (28 days- | | | | |
| | 23 months) | | | | |
| | Children (2-11 years) | | | | |
| | Adolescents (12-17 years) | | | | |
| | Adults (18-64 years) | | | | |
| | From 65-84 years | | | | |
| | 85 years and over | | | | |
| | Missing | | | | |

Gr 1 = Group 1 description

N = number of subjects

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories Missing = <describe missing>

### Template 24 Number of subjects by country

| | ACWY-TT | ACWYHPV | HPV | Co-ad | Tdap | Total |
|---|---|---|---|---|---|---|
| | N = 259 | N = 259 | N = 261 | N = 260 | N = 261 | N = 1300 |
| Country | n | n | N | n | n | n |
| Dominican Republic | 86 | 87 | 88 | 87 | 87 | 435 |
| Estonia | 87 | 86 | 87 | 87 | 88 | 435 |
| Thailand | 86 | 86 | 86 | 86 | 86 | 430 |

ACWY-TT = Subjects who received MenACWY-TT at Month 0 and Cervarix at Month 1, 2 and 7

ACWYHPV = Subjects who received MenACWY-TT and Cervarix at Month 0 and Cervarix at Month 1 and 6 HPV = Subjects who received Cervarix at Month 0, 1 and 6

Co-ad = Subjects who received MenACWY-TT, Cervarix and Boostrix at Month 0 and Cervarix at Month 1 and 6 Tdap = Subjects who received Boostrix and Cervarix at Month 0 and Cervarix at Month 1 and 6

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories

## Template 25 Listing of dropouts due to AEs, SAEs and solicited symptoms (Total cohort)

| Study-<br>Subject<br>No. | Country | Gender | AE Description | SAE | Causality | Outcome | Type of discontinuation |
|---|---|---|---|---|---|---|---|
| PP<br>D | Germany | F | SUBJECT DIED | Y | | Fatal | Study at visit/contact: VISIT11 (Y5) |
| PP<br>D | Germany | F | SUBJECT DIED | Υ | | Fatal | Study at visit/contact: VISIT11 (Y5) |

Gr 2 = Group 2 description

Gr 3 = Group 3 description

N = Number of enrolled subjects

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Final

## Template 26 Percentage of subjects with large injection site reaction during the 4-day (Days 0-3) period after Boostrix (Total Vaccinated Cohort)

| Type of Swelling | (Each group)<br>N= | | | | Total<br>N= | | | |
|---|---|---|---|---|---|---|---|---|
| | n | % 95%CI | | n | % | 95% CI | | |
| | | | LL | UL | | | LL | UL |
| Any | | | | | | | | |
| Local Swelling | | | | | | | | |
| Diffuse Swelling | | | | | | | | |
| Involving at least one adjacent | | | | | | | | |
| joint | | | | | | | | |

Boostrix group= Subjects who had received GSK Biologicals' Tdap vaccine (Boostrix) in study 106316 and a second dose of Tdap vaccine (Boostrix) at Year 9 Visit 6

Adacel group= Subjects who had received Sanofi Pasteurs' Tdap vaccine (Adacel) in study 106316 and a second dose of Tdap vaccine (Boostrix) at Year 9 Visit 6

Control group= Subjects who will receive the first dose of Tdap vaccine (Boostrix) at Year 9 Visit 6

N = Number of subjects with documented dose

n/% = number/percentage of subjects reporting a specified symptom

95% CI = Standardized asymptotic 95% confidence interval, LL = Lower Limit, UL = Upper Limit

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

| Statistical Analysis Plan |
|---|
| A phase III, open-label, single-group, multi-centre study to assess the immunogenicity, safety and reactogenicity of GSK Biologicals' combined reduced antigen content diphtheria, tetanus and acellular pertussis (dTpa) vaccine, <i>Boostrix</i> , administered as a booster dose in healthy Russian subjects aged four years and older. |
| 201532 [DTPA (BOOSTRIX)-050] |
| All analyses as planned per protocol and for study report. |
| Amendment 1 Final: 10 March 2019 |
| (Lead Statistician) |
| PPD (Study statistician) |
| R&D Project Leader) (Clinical and Epidemiology |
| , Clinical Research and Development Lead (CRDL) |
| (Study statistician) |
| (peer reviewer statistician) |
| (public disclosure) |
| (Scientific writer) |
| (Lead statistical analyst) |
| (Global Regulatory Affairs) |
| PPD and PPD (Safety Physician) |

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

| | Statistical Analysis Plan Amendment 1 Final |
|---|---|
| Amendment 1 reviewed by: | Project Leader) (Clinical and Epidemiology R&D |
| | PPD , Clinical Research and Development Lead (CRDL) |
| | (Lead statistician) |
| | (Scientific writer) |
| | (Lead stat analyst) |
| Approved by: | PPD (Clinical and Epidemiology R&D Project Leader) |
| | PPD , Clinical Research and Development Lead (CRDL) |
| | (Study statistician) |
| | (Lead Statistician) |
| | PPD (Lead stat analyst, approver) |
| | (Scientific writer) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 14April 2017)

## 201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| LIS | ST OF A | ABBREVIATIONS | 8 |
| 1. | DOC | JMENT HISTORY | 10 |
| 2. | STUE | DY DESIGN | 10 |
| 3. | OBJE | CTIVES | 12 |
| Ο. | 3.1. | Primary objectives | |
| | 3.2. | Secondary objectives | |
| 4. | ENDF | POINTS | 12 |
| • | 4.1. | Primary endpoints | |
| | 4.2. | Secondary endpoints | |
| 5. | ANAL | YSIS SETS | 14 |
| | 5.1. | Definition | |
| | | 5.1.1. Total vaccinated cohort (TVC) | |
| | | 5.1.2. Per protocol cohort for analysis of immunogenicity | 14 |
| | 5.2. | Criteria for eliminating data from Analysis Sets | 15 |
| | | 5.2.1. Elimination from Total vaccinated cohort (TVC) | 15 |
| | | 5.2.2. Elimination from ATP cohort for immunogenicity | 16 |
| | | 5.2.2.1. Excluded subjects | |
| | | 5.2.2.2. Right censored Data | 17 |
| | | 5.2.2.3. Visit-specific censored Data | 17 |
| | 5.3. | Important protocol deviation not leading to elimination from ATP cohort for immunogenicity | 17 |
| 6. | STAT | ISTICAL ANALYSES | |
| | 6.1. | Demography | |
| | | 6.1.1. Analysis of demographics/baseline characteristics planned | |
| | | in the protocol | |
| | | 6.1.2. Additional considerations | |
| | 6.2. | Exposure | |
| | | 6.2.1. Analysis of exposure planned in the protocol | |
| | 0.0 | 6.2.2. Additional considerations | |
| | 6.3. | Immunogenicity | |
| | | 6.3.1. Analysis of immunogenicity planned in the protocol | |
| | 0.4 | 6.3.2. Additional considerations | |
| | 6.4. | Analysis of safety | |
| | | 6.4.1. Analysis of safety planned in the protocol | |
| | | 6.4.2. Additional considerations | 22 |
| 7. | ANAL | YSIS INTERPRETATION | <mark>22</mark> |
| 8. | | DUCT OF ANALYSES | |
| | 8.1. | Sequence of analyses | |
| | 8.2. | Statistical considerations for interim analyses | |
| | 8.3. | Statistical considerations for interim analyses | 23 |

| | | | | Statistical Analysis Plan Amendmen | |
|---|---|---|---|---|---|
| 9. | CHAN | GES FRO | OM PLANNED ANALYSES | | 23 |
| 10. | LIST | F FINAL | REPORT TABLES, LISTING | GS AND FIGURES | 24 |
| 11. | | | IDARD DATA DERIVATION | RULE AND STATISTICAL | 24 |
| | 11.1. | Statistica<br>Standard<br>11.2.1.<br>11.2.2.<br>11.2.3. | al Method Referencesd data derivation Date derivation Demography Immunogenicity | | 24<br>25<br>25<br>25 |
| 12. | ANNE | | • | ODES | |
| 13 | ΔNNE | X 3. STH | DV SPECIFIC MOCK TEI | | 30 |

## 201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

## **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Study group and epoch foreseen in the study | 11 |
| Table 2 | Study group and treatment foreseen in the study | 11 |
| Table 3 | Blinding of study epoch | 11 |
| Table 4 | Age stratification | 18 |
| Table 5 | Humoral Immunity (Antibody determination) | 20 |
| Table 6 | Intensity scales to be used by the parent(s)/LAR(s) for solicited symptoms during the solicited follow-up period | 27 |
| Table 7 | Intensity scales for solicited symptoms in adults and children of six years of age or more | 28 |

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

## **LIST OF TEMPLATES**

| | PAGE |
|---|---|
| Template 1 | Number of subjects enrolled by center (Total Vaccinated Cohort)30 |
| Template 2 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal at Visit 3 (Total Vaccinated Cohort) |
| Template 3 | Number of subjects at each visit and list of withdrawn subjects (Total Vaccinated Cohort) |
| Template 4 | Number of subjects enrolled into the study as well as the number of subjects excluded from ATP analyses with reasons for exclusion |
| Template 5 | Deviations from specifications for age and intervals between study visits (Total Vaccinated Cohort) |
| Template 6 | Summary of demographic characteristics (ATP cohort for Immunogenicity) |
| Template 7 | Summary of vital signs characteristics (Total Vaccinated Cohort)34 |
| Template 8 | Study population (Total Vaccinated Cohort)34 |
| Template 9 | Seropositivity and seroprotection rates and GMCs for anti-<br>diphtheria and anti-tetanus antibodies before and one month<br>after the booster vaccination (ATP cohort for immunogenicity)35 |
| Template 10 | Booster responses for anti-PT, anti-FHA and anti-PRN antibody concentration one month after the booster vaccination (ATP cohort for immunogenicity) |
| Template 11 | Reverse cumulative curve for anti-diphtheria antibody concentration one month after the booster vaccination (ATP cohort for immunogenicity) |
| Template 12 | Seroprotection rate for anti-Diphtheria antibody concentration by ELISA and VERO NEUTRALISATION (ATP cohort) |
| Template 13 | Compliance in returning symptom information (Total Vaccinated Cohort) |
| Template 14 | Incidence and nature of grade 3 symptoms (solicited and unsolicited) reported during the 4-day (Days 0-3) period after vaccination following each dose and overall (Total Vaccinated Cohort) |
| Template 15 | Incidence of solicited local symptoms reported during the 4-day (Days 0-3) period after vaccination following each dose and overall (Total Vaccinated Cohort) |

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final Incidence of solicited general symptoms reported during the 4-Template 16 day (Days 0-3) post-vaccination period (Total Vaccinated Cohort) .......40 Template 17 Percentage of subjects with grade 3 unsolicited symptoms classified by MedDRA SOC and PT from Day 0 to Day 30 after any vaccination (Total Vaccinated Cohort) ......41 Template 18 Number (%) of subjects with serious adverse events from first study vaccination up to Visit 3 including number of events reported (Total Vaccinated Cohort) ......43 Subjects with Serious Adverse Events reported up to Visit 2 Template 19 (Total Vaccinated Cohort) ......44 Template 20 Number and percentage of subjects who started at least one concomitant medication from Day 0 to Day 7 (Total Vaccinated Solicited and Unsolicited symptoms experienced by subjects Template 21 classified by MedDRA Primary System Organ Class and Preferred Term within the 31-day (Days 0-30) post-vaccination period - SAE excluded (Total vaccinated cohort)......46 Template 22 Minimum and maximum activity dates (TVC) .......46 Template 23 Number of enrolled subjects by age category (TVC) .......47 Template 24 Number of subjects by country......47 Template 25 Listing of dropouts due to AEs, SAEs and solicited symptoms Template 26 Percentage of subjects with large injection site reaction during the 4-day (Days 0-3) period after Boostrix (Total Vaccinated Template 27 GMCs fold increase for anti-D, anti-T, anti-PT, anti-FHA and anti-PRN antibodies one month after the booster vaccination by study

(Per protocol cohort for analysis of immunogenicity) .......48

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

#### LIST OF ABBREVIATIONS

AE Adverse event

ANOVA Analysis of Variance

ATP Per Protocol Set

BS Blood Sample

cDISCI Clinical Data Interchange Standards Consortium

CI Confidence Interval

CRF Case Report Form

CTRS Clinical Trial Registry Summary

EL.U/ml ELISA unit per milliliter

Eli Type Internal GSK database code for type of elimination code

ELISA Enzyme-linked immunosorbent assay

GE Gastroenteritis

GSK GlaxoSmithKline

iDMC Independent Data Monitoring Committee

IU/ml International units per milliliter

LL Lower Limit of the confidence interval

MedDRA Medical Dictionary for Regulatory Activities

N.A. Not Applicable

PD Protocol Deviation

SAE Serious adverse event

SAP Statistical Analysis Plan

SAS Statistical Analysis Software

SBIR GSK Biological's Internet Randomization System

SD Standard Deviation

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

SR Study Report

TFL Tables Figures and Listings

TOC Table of Content

TVC Total Vaccinated Cohort

UL Upper Limit of the confidence interval

#### 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|---------------|-----------------------------------|
| 09-OCT-2017 | first version | Amendment 02 Final 1: 07-AUG-2017 |
| 10-MAR-2019 | Amendment 1* | Amendment 02 Final 1: 07-AUG-2017 |

<sup>\*</sup> summary of GMC fold increase from pre to post vaccination has been added.

#### 2. STUDY DESIGN

<u>Visit:</u> <u>Visit 1</u> <u>Visit 2</u>

<u>Timepoint:</u> Day 1 Day 31

Blood sampling: Pre-Booster Post-Booster

Vaccination Study End

Age: ≥ 4 yrs

Protocol waivers or exemptions are not allowed unless necessary for the management of immediate safety concerns. Therefore, adherence to the study design requirements, including those specified in the outline of study procedures (Section 5.5 of the protocol), are essential and required for study conduct.

- Experimental design: Phase III, open-label, non-randomised, multi-centric, single-country study with a single group.
- Duration of the study:
  - Epoch 001: Primary Epoch starting at Visit 1 (Day 1) and ending at Visit 2 (Day 31)
- Primary Completion Date (PCD): Visit 2 (Day 31)
- End of Study (EoS): Last testing results released of samples collected at Visit 2.
- Study groups: The study group and epoch foreseen in this study is presented in Table 1.

<sup>\*</sup> An equal number of subjects are expected to be recruited in the following age categories: 4-9 years (children), 10-17 years (adolescents), 18-64 years (adults) and ≥65 years (elderly population) in order to evaluate data.

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

Table 1 Study group and epoch foreseen in the study

| Study group | Number of | Age (Min) | Epoch |
|-------------|-----------|-----------|-----------|
| Study group | subjects | | Epoch 001 |
| dTpa Group | 448 | ≥4 years | X |

#### Table 2 Study group and treatment foreseen in the study

| Treatment name | Vaccine/Product name | Study Group |
|----------------|-----------------------|-------------|
| Treatment name | Vaccine/i Todact name | dTpa Group |
| Boostrix | dTpa | X |

- Control: uncontrolled (in terms of no active comparator).
- Vaccination schedule: A single dose of *Boostrix* vaccine will be administered to all subjects at Visit 1 (Day 1).
- Treatment allocation: Non-randomised and stratified by age.
- Blinding: open.

Table 3 Blinding of study epoch

| Study Epoch | Blinding |
|-------------|----------|
| Epoch 001 | open |

- Sampling schedule: A blood sample of approximately 5 ml will be collected from all subjects before vaccination (at the Pre-Booster timepoint) and one month after vaccination (Post-Booster timepoint).
- Type of study: self-contained.
- Data collection: Electronic Case Report Form (eCRF).

#### 3. OBJECTIVES

## 3.1. Primary objectives

• To assess the immune response to the dTpa vaccine in terms of seroprotection status for antibodies against diphtheria and tetanus antigens and in terms of seropositivity status for antibodies against the pertussis antigens [pertussis toxoid (PT), filamentous haemagglutinin (FHA) and pertactin (PRN)], one month after vaccination.

Refer to Section 4.1 for the definition of the primary endpoints.

## 3.2. Secondary objectives

- To assess the immune response in terms of booster response\* to diphtheria, tetanus, PT, FHA, and PRN antigens, one month after vaccination.
- To assess the immune response in terms of antibody concentrations to diphtheria, tetanus, PT, FHA, and PRN antigens, one month after vaccination.
- To assess the reactogenicity and safety of Boostrix in terms of solicited symptoms (local and general), unsolicited adverse events (AEs) and serious adverse events (SAEs).

Refer to Section 4.2 for the definition of the secondary endpoints.

#### 4. ENDPOINTS

## 4.1. Primary endpoints

- Immunogenicity with respect to components of the study vaccine.
  - Anti-diphtheria\* and anti-tetanus seroprotection status (ie antibody concentrations ≥0.1 IU/ml), one month after vaccination.
  - Anti-PT, anti-FHA and anti-PRN seropositivity status (ie antibody concentration is greater than or equal to the assay cut-off value), one month after vaccination.

## 4.2. Secondary endpoints

- Booster response to the diphtheria, tetanus and pertussis (PT, FHA and PRN) antigens, one month after vaccination.
  - Booster response to Diphtheria and Tetanus antigens is defined as:
    - o for subjects with pre-vaccination antibody concentration <0.1 IU/ml (i.e. below the seroprotection cut-off), antibody concentrations at least ≥0.4 IU/ml, one month after vaccination, and

<sup>\*</sup>Sera with ELISA concentrations <0.1 IU/ml will be tested for neutralising antibodies using a Vero-cell neutralisation assay.

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

- o for subjects with pre-vaccination antibody concentration ≥0.1 IU/ml (i.e. equal or above the seroprotection cut-off), an increase in antibody concentrations of at least four times the pre-vaccination concentration, one month after vaccination
- Booster response to PT, FHA and PRN antigens is defined as:
  - o for subjects with pre-vaccination antibody concentration below the assay cut-off, post-vaccination antibody concentration ≥ four times the assay cut-off,
  - o for subjects with pre-vaccination antibody concentration between the assay cut-off and below four times the assay cut-off, post-vaccination antibody concentration ≥ four times the pre-vaccination antibody concentration, and
  - o for subjects with pre-vaccination antibody concentration ≥ four times the assay cut-off, post-vaccination antibody concentration ≥ two times the pre-vaccination antibody concentration
- Immunogenicity with respect to components of the study vaccine.
  - Anti-diphtheria anti-tetanus, anti-PT, anti-FHA and anti-PRN antibody concentrations, one month after vaccination.
- Solicited local and general symptoms.
  - Occurrence of each solicited local and general symptom during the 4-day (Day 1-4) follow-up period after vaccination.
  - Occurrence of large swelling reactions during the 4-day (Day 1-4) follow-up period after vaccination.
- Unsolicited adverse events.
  - Occurrence of unsolicited AEs during the 31-day (Day 1-31) follow-up period after vaccination, according to the Medical Dictionary for Regulatory Activities (MedDRA) classification.
- Serious adverse events.
  - Occurrence of SAEs from the vaccination up to study end.

#### 5. ANALYSIS SETS

#### 5.1. Definition

## 5.1.1. Total vaccinated cohort (TVC)

The TVC will include all subjects with at least one study vaccine administration documented.

- A safety analysis based on the TVC will include all vaccinated subjects.
- An immunogenicity analysis based on the TVC will include all vaccinated subjects for whom immunogenicity data are available.

Note that enrolled subjects who gave informed consent or blood sample pre-vaccination but were not vaccinated will be excluded from TVC.

## 5.1.2. Per protocol cohort for analysis of immunogenicity

The PP cohort for immunogenicity will include all evaluable subjects:

- Who have received the dose of study vaccine.
- For whom administration site of study vaccine is known and according to the protocol.
- Who have not received a vaccine not specified or forbidden in the protocol.
- Who meet all eligibility criteria.
- Who are within the maximum interval (the interval between Visit 1 and blood sampling at Visit 2, considered for inclusion of a subject will be 21–48 days) allowed as defined in the protocol.
- Who did not receive a product leading to exclusion from a PP analysis (refer to Section 6.7.2 of the protocol, namely
  - Any investigational or non-registered product (drug or vaccine) other than the study vaccine used during the study period.
  - Immunosuppressants or other immune-modifying drugs administered chronically (i.e. more than 14 days) during the study period. For corticosteroids, this will mean prednisone ≥20 mg/day (for adult subjects) or ≥0.5 mg/kg/day (for paediatric subjects), or equivalent. Inhaled and topical steroids are allowed.
  - Long-acting immune-modifying drugs administered at any time during the study period (e.g. infliximab).
  - A vaccine not foreseen by the study protocol administered during the period starting from the dose of study vaccine (Day 1) and ending 31 days after the dose of vaccine administration, with the exception of influenza vaccine which is allowed throughout the study period.

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

- In case an emergency mass vaccination for an unforeseen public health threat (e.g.: a pandemic) is organised by the public health authorities, outside the routine immunisation program, the time period described above can be reduced if necessary for that vaccine provided it is licensed and used according to its Summary of Product Characteristics (SmPC) and according to the local governmental recommendations and provided a written approval of the Sponsor is obtained.
- Immunoglobulins and/or any blood products administered during the study period.)
- Who did not present with a medical condition leading to exclusion from an PP analysis (refer to Section 6.8 of the protocol, namely subjects will be eliminated from the PP cohort for immunogenicity if, during the study, they incur a condition that has the capability of altering their immune response or are confirmed to have an alteration of their initial immune status).
- For whom data concerning immunogenicity endpoint measures are available post vaccination. This will include subjects for whom assay results are available for antibodies against at least one study vaccine antigen component.

## 5.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each sets.

### 5.2.1. Elimination from Total vaccinated cohort (TVC)

Code 1030 (Study vaccine not administered at all) and code 900 (invalid informed consent or fraud data) will be used for identifying subjects eliminated from TVC.

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

## 5.2.2. Elimination from ATP cohort for immunogenicity

## 5.2.2.1. Excluded subjects

A subject will be excluded from the ATP cohort for immunogenicity under the following conditions

| Code | Decode => Condition under which the code is used |
|---|---|
| 900 | Questionable subject => Invalid informed consent or fraudulent data. In case informed consent is obtained retrospectively the subject is not eliminated. |
| 1030 | Study vaccine dose not administrated at all but subject number allocated => subjects enrolled but not vaccinated |
| 1040 | Administration of vaccine(s) forbidden in the protocol => |
| | Any investigational or non-registered product (drug or vaccine) other than the study vaccine used during the study period. |
| | • A vaccine not foreseen by the study protocol administered during the period starting from the dose of study vaccine (Day 1) and ending 31 days after the dose of vaccine administration, with the exception of influenza vaccine which is allowed throughout the study period. This includes emergency mass vaccination for an unforeseen public health threat (e.g.: a pandemic) organised by the public health authorities, outside the routine immunisation program. |
| 1070 | Study vaccine dose not administered according to protocol => for instance • Route of vaccination is not Intramuscular for Boostrix |
| | <ul> <li>Wrong reconstitution of Boostrix before injection</li> </ul> |
| 1080 | Vaccine temperature deviation => Boostrix vaccine administered despite a Good Manufacturing Practices (GMP) no-go temperature deviation |
| 1090 | Expired vaccine administered=> Subjects who received an expired Boostrix vaccine |
| 2010 | Protocol violation (inclusion/exclusion criteria) => ineligible subject: • age below (excluding) 4 year |
| | • Other considerations as stated in section 4.2 – 4.3 in the protocol |

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

| 2040 | Administration of any medication forbidden by the protocol=> |
|---|---|
| 2040 | • Administration of any medication forbidden by the protocol=> |
| | <ul> <li>Immunosuppressants or other immune-modifying drugs administered chronically (i.e. more than 14 days) during the study period. For corticosteroids, this will mean prednisone ≥20 mg/day (for adult subjects) or ≥0.5 mg/kg/day (for paediatric subjects), or equivalent. Inhaled and topical steroids are allowed.</li> </ul> |
| | <ul> <li>Long-acting immune-modifying drugs administered at any<br/>time during the study period (e.g. infliximab).</li> </ul> |
| | <ul> <li>Immunoglobulins and/or any blood products administered during the study period.)</li> </ul> |
| 2070 | Concomitant infection not related to the vaccine which may influence immune response = > subject who incurs a condition that has the capability of altering their immune response or are confirmed to have an alteration of their initial immune status |
| 2090 | Non-compliance with the blood sampling schedule (including wrong and unknown dates) => Blood sample not collected within 21 days-48 days after the Boostrix vaccine. |
| 2100 | Essential serological data missing => No serological results at all available post-vaccination (Visit 2) |
| 2120 | Obvious incoherence or abnormality or error in data => • BS result available while BS not taken |
| | <ul> <li>Post vaccination results below pre-vaccination results for all<br/>available assays tested at pre-vaccination ie PT, FHA, PRN,<br/>Diphtheria (ELISA), Tetanus</li> </ul> |

## 5.2.2.2. Right censored Data

Not applicable

## 5.2.2.3. Visit-specific censored Data

Not applicable

## 5.3. Important protocol deviation not leading to elimination from ATP cohort for immunogenicity

Refer to the protocol deviaito management plan for important protocol deviation not leading to elimination from ATP cohort for immunogenicity.

#### 6. STATISTICAL ANALYSES

Note that standard data derivation rule and stat methods are described in section 11 and will not be repeated below.

## 6.1. Demography

## 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

Demographic characteristics (age at vaccination visit in years, gender and geographical ancestry, body mass index in kg/m<sup>2</sup>), cohort description and withdrawal status will be summarised using descriptive statistics:

- Frequency tables will be generated for categorical variable such as centre.
- Mean, median, standard deviation will be provided for continuous data such as age.
- The distribution of subjects based on age stratification will be tabulated (as seen in Table 4).

In addition, the above analysis will also be done for sub-groups based on age as an exploratory analysis.

Table 4 Age stratification

| Age groups | Number of subjects |
|-------------|--------------------|
| 4-9 years | ~112 |
| 10-17 years | ~112 |
| 18-64 years | ~112 |
| ≥65 years | ~112 |

#### 6.1.2. Additional considerations

All demography summaries will be generated for the TVC and ATP cohort. An additional age split will be added in the 4-9 years group to determine the distribution of subjects below 6 year old as solicited symptoms are different (see section 11.2.4).

Number and reason for elimination from ATP will be tabulated.

## 6.2. Exposure

## 6.2.1. Analysis of exposure planned in the protocol

Not described in the protocol as a single dose is provided and the number of vaccinated subjects is provided.

#### 6.2.2. Additional considerations

Not applicable.

### 6.3. Immunogenicity

#### 6.3.1. Analysis of immunogenicity planned in the protocol

The primary analysis will be based on the PP cohort for analysis of immunogenicity. If, the percentage of vaccinated subjects with serological results excluded from the PP cohort for analysis of immunogenicity is 5% or more, a second analysis based on the TVC will be performed to complement the PP analysis.

For all subjects and each antigen:

- Seropositivity/seroprotection rate at pre-vaccination and one month post-vaccination will be calculated with exact 95% CIs.
- GMCs at pre-vaccination and one month post-vaccination will be tabulated with 95% CIs.
- Booster response rate one month post-vaccination will be calculated with exact 95% CIs for diphtheria, tetanus and pertussis antigens.

In addition, the above analysis will also be done based on age stratification (Refer Table 4) as an exploratory analysis.

Finally, antibody concentrations distribution at pre-vaccination and one month post-vaccination will be displayed using reverse cumulative curves (RCC).

#### Handling of missing data:

• For a given subject and a given immunogenicity measurement, missing or nonevaluable measurements will not be replaced. Therefore, an analysis will exclude subjects with missing or non-evaluable measurements.

#### 6.3.2. Additional considerations

Increase in GMC from pre-vaccination to post-vaccination will be computed with 95% CI.

Seroprotection and booster response is defined in section 4. The percentage of subjects with ELISA anti-Diphtheria above 0.1 IU/ml or with Vero anti-Diphtheria above 0.01 IU/ml will be summarized at pre and post vaccination. In case subjects with ELISA anti-Diphtheria above 0.1 IU/ml have no result by Vero, the subjects will be treated as censored for Vero anti-Diphtheria and survival method will be used to estimate percentage and associated CI.

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

A seronegative subject is a subject whose antibody concentration is below the assay cutoff value. A seropositive subject is a subject whose antibody concentration is greater than or equal to the assay cut-off value.

The thresholds defining seropositivity are provided below

Table 5 Humoral Immunity (Antibody determination)

| System | Component | Method | Kit/Manufacturer | Unit | Cut-off <sup>†</sup> | Laboratory* |
|---|---|---|---|---|---|---|
| Serum | Corynebacterium<br>diphtheriae.Diphtheria<br>Toxoid Ab.IgG | ELI | NA | IU/ml | 0.057 | GSK Biologicals or designated laboratory |
| Serum | Corynebacterium<br>diphtheriae.Diphtheria<br>Toxoid Ab | NEU<br>assay on<br>Vero<br>cells** | NA | IU/ml | 0.004 | GSK Biologicals<br>or designated<br>laboratory |
| Serum | Clostridium<br>tetani.Tetanus Toxoid<br>Ab.IgG | ELI | NA | IU/ml | 0.043 | GSK Biologicals or designated laboratory |
| Serum | Bordetella<br>pertussis.Pertussis<br>Toxin Ab.IgG | ELI | NA | IU/ml | 2.693 | GSK Biologicals or designated laboratory |
| Serum | Bordetella<br>pertussis.Filamentous<br>Hemaglutinin Ab.lgG | ELI | NA | IU/ml | 2.046 | GSK Biologicals<br>or designated<br>laboratory |
| Serum | Bordetella<br>pertussis.Pertactin<br>Ab.IgG | ELI | NA | IU/ml | 2.187 | GSK Biologicals<br>or designated<br>laboratory |

ELI: ELISA

NEU: Neutralisation assay

NA: Not Applicable

IU/ml: International Units per millilitre

<sup>†</sup>Assays for diphtheria, tetanus and pertussis were re-developed and re-validated as per most recent CBER recommendations (Guidance for Industry "Bioanalytical Method Validation" from September 2013). The new assay cutoff's that apply are listed in the table.

<sup>\*</sup>GSK Biologicals laboratory refers to the Clinical Laboratory Sciences (CLS) in Rixensart, Belgium and Wavre, Belgium.

<sup>\*\*</sup>Test on Vero-cells will be performed on pre- and post-vaccination samples with concentrations <0.1 IU/ml by ELISA.

## 6.4. Analysis of safety

### 6.4.1. Analysis of safety planned in the protocol

The analysis will be based on the TVC.

- The percentage of subjects reporting each individual solicited local and general symptom during the 4-day (Day 1-4) follow-up period after booster vaccination will be tabulated. The same calculations will be done for each individual solicited symptom rated as grade 3 in intensity and for each individual solicited symptom assessed as causally related to vaccination.
- Occurrence of fever during the 4-day follow-up period after vaccination will be reported per 0.5°C cumulative increments.
  - In addition, the above analysis will also be done for sub groups based on age stratification (Refer Table 4) as an exploratory analysis.
- The percentage of subjects with at least one local symptom (solicited or unsolicited), with at least one general symptom (solicited or unsolicited) and with any symptom (solicited or unsolicited) during the 4-day (Day 1-4) follow-up period after booster vaccination will be tabulated with exact 95% CI after booster vaccination. The same calculations will be done for symptoms (solicited or unsolicited) rated as grade 3 in intensity, for symptoms (solicited or unsolicited) leading to medical consultation and for symptoms (solicited or unsolicited) assessed as causally related to vaccination.
- The percentage of subjects who started to receive at least one concomitant medication (i.e. any medication, antipyretic medication, prophylactic antipyretics) during the 4-day (Day 1-4) and 31-day (Day 1-31) follow-up period after vaccination will be tabulated with exact 95% CI.
- The verbatim reports of unsolicited AEs will be reviewed by a clinical research and development lead and the signs and symptoms will be coded according to MedDRA. Every verbatim term will be matched with the appropriate Preferred Term. The percentage of subjects with unsolicited AEs occurring within the 31-day (Day 1-31) follow-up period after booster dose with its exact 95% CI will be tabulated by Preferred Term. Similar tabulation will be done for unsolicited AEs rated as grade 3 and for unsolicited AEs with causal relationship to vaccination.
- Any large injection site reaction (for subjects <6 years of age defined as a swelling with a diameter of >50 mm and for subjects ≥6 years of age swelling with a diameter of >100 mm, noticeable diffuse swelling or noticeable increase in limb circumference) onset during the 4-day (Day 1-4) follow-up period after vaccination will be described in detail.
- SAEs and withdrawal due to AEs and SAEs will be described in detail.

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

#### Handling of missing data:

- For a given subject and the analysis of solicited symptoms four days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore the analysis of the solicited symptoms based on the TVC will include only vaccinated subjects and doses with documented safety data (i.e., symptom screen completed).
- For analysis of unsolicited AEs, such as SAEs or AEs by primary Medical Dictionary for Regulatory Activities (MedDRA) term, and for the analysis of concomitant medications, all vaccinated subjects will be considered. Subjects, who do not report the event or the concomitant medication, will be considered as subjects without the event or the concomitant medication, respectively.
- For summaries reporting both solicited symptoms and unsolicited AEs, all vaccinated subjects will be considered. Subjects, who do not report the event or the concomitant medication, will be considered as subjects without the event or the concomitant medication, respectively.

#### 6.4.2. Additional considerations

The summary of each solicited symptoms and unsolicited adverse event will also be done for medically attended symptom/adverse event and for grade 3 causally related AE.

### 7. ANALYSIS INTERPRETATION

All analyses will be conducted in a descriptive manner.

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

## 8. CONDUCT OF ANALYSES

Any deviation(s) or change(s) from the original statistical plan outlined in this protocol will be described and justified in the final study report.

## 8.1. Sequence of analyses

Analysis of the single booster dose will be performed at the end of the study when all data are available. An integrated clinical study report containing all data will be written and made available to the investigators.

## 8.2. Statistical considerations for interim analyses

All analyses will be conducted on final data and therefore no statistical adjustment for interim analyses is required.

| Description | Analysis<br>ID | Disclosure Purpose (IN=internal, CTRS=public posting, SR=study report and public posting) | Dry run<br>review<br>needed (Y/N) | Study Headline Summary (SHS)requiring expedited communication to upper management (Yes/No) | Reference for TFL |
|---|---|---|---|---|---|
| Final | E1 01 | SR | Yes | Yes | TFL TOC |

## 8.3. Statistical considerations for interim analyses

Not applicable

#### 9. CHANGES FROM PLANNED ANALYSES

Template 27 is a new addition to the SAP as per the dry run meeting minutes.

As per the dry run meeting minutes the TFL TOC is update by adding few additional tables, and more details are available in the dry run meeting minutes. Below is the link to refer to the dry run meeting minutes in eTMF

https://biodocumentum.bio.corpnet1.com/webtoppr/drl/objectId/090f45f688621990

Few tables were split as two separate tables in the updated TFL TOC by age category (as <6 years and  $\ge 6$  years), as the intensity score for the solicited symptoms are different for both the age categories.

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

## 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The TFL TOC provides the list of tables/listings and figures needed for the study report. It also identifies the tables eligible for each analysis and their role (synopsis, in-text, post-text, SHS, CTRS,...). Note that all TFL aimed to be included as post-text are noted as post-text even if these are tabulation of individual data such as listing of SAE. The post-text material contains all source material for the study report and accordingly a post-text table may be redundant with an in-text table.

The mock tables referred under column named 'layout' can be found in section 13 of this SAP.

The following group name will be used in the TFLs, to be in line with the T-domains:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | dTpa Group | Boostrix |

## 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS

#### 11.1. Statistical Method References

The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413].

If some samples with anti-D concentrations < 0.1 IU/mL cannot be retested by VERO, VERO will be treated as left censored at 0.1 IU/mL and the Greenwoood formula for censored data will be used to estimate the percentage of subjects with anti-D antibody concentrations  $\geq$ 0.1 IU/mL by ELISA or anti-D concentrations  $\geq$ 0.01 IU/mL by VERO and its associated CI.

The 95% CI for GMTs/GMCs will be obtained within each group separately. The 95% CI for the mean of log-transformed titre/concentration will be first obtained assuming that log-transformed values were normally distributed with unknown variance. The 95% CI for the GMTs/GMCs will then be obtained by exponential-transformation of the 95% CI for the mean of log-transformed titre/concentration.

#### 11.2. Standard data derivation

#### 11.2.1. Date derivation

- SAS date derived from a character date: in case day is missing, 15 is used. In case day & month are missing, 30June is used.
- Onset day for an event (AE, medication, vaccination, ...): the onset day is the number of days between the last study vaccination & the onset/start date of the event. This is 0 for an event starting on the same day as a vaccination. See SAS date derived in case the start date of the event is incomplete.

## 11.2.2. Demography

Age: Age at the reference activity, computed as the number of complete weeks between the date of birth and the reference activity.

Conversion of weight to kg: the following conversion rule is used:

Weight in Kilogram= weight in Pounds / 2.2 + weight in ounces / 35.2

The result is rounded to 2 decimals.

Conversion of height to cm: the following conversion rule is used:

Height in Centimetres = Height in Feet \* 30.48+

Height in Inch \* 2.54

The result is rounded to the unit (ie no decimal).

Conversion of temperature to °C: the following conversion rule is used:

Temperature in °Celsius = ((Temperature in °Fahrenheit -32) \*5)/9

The result is rounded to 1 decimal.

## 11.2.3. Immunogenicity

• The geometric mean titres (GMTs)/geometric mean concentrations (GMCs) calculations will be performed by taking the anti-log of the mean of the log10 titre/concentration transformations. Antibody titres/concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off for the purpose of GMT/GMC calculation.

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

- In general, the assay cut-off is the value under which there is no quantifiable result available. For an assay with a specific 'assay cut\_off', numerical immuno result is derived from a character field (rawres):
  - If rawres is 'NEG' or '-' or '(-)', numeric result= assay cut\_off/2,
  - if rawres is 'POS' or '+' or '(+)', numeric result = assay cut off,
  - if rawres is '< value' and value<=assay cut off, numeric result =assay cut off/2,</li>
  - if rawres is '< value' and value>assay cut off, numeric result =value,
  - if rawres is '> value' and value<assay cut\_off, numeric result =assay cut\_off/2,
  - if rawres is '> value' and value>=assay cut off, numeric result =value,
  - if rawres is '<= value' or '>= value' and value<assay cut\_off, numeric result =assay cut\_off/2,</p>
  - if rawres is '<= value' or '>= value' and value>=assay cut\_off, numeric result
     =value,
  - if rawres is a value < assay cut off, numeric result = assay cut off/2,</li>
  - if rawres is a value >= assay cut off, numeric result = rawres,
  - else numeric result is left blank

#### 11.2.4. Safety

For analysis of solicited, unsolicited adverse events (such as serious adverse events or adverse events by primary MedDRA term) and for the analysis of concomitant medications, all vaccinated subjects will be considered. Subjects who did not report the event or the concomitant medication will be considered as subjects without the event or the concomitant medication respectively.

The following rules will be used for the analysis of solicited symptoms:

- Subjects who documented the absence of a solicited symptom will be considered not having that symptom.
- Subjects who documented the presence of a solicited symptom and fully or partially recorded daily measurement over the solicited period will be included in the summaries at that dose and classified according to their maximum observed daily recording over the solicited period.
- Subjects who documented the presence of a solicited symptom without having recorded any daily measurement will be considered as having that symptom (at the lowest intensity).
- Intensity of the following solicited AEs will be assessed as described in Table 6 and below
201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

Table 6 Intensity scales to be used by the parent(s)/LAR(s) for solicited symptoms during the solicited follow-up period

| Toddler/Child (<6 years) | | |
|---|---|---|
| Adverse Event | Intensity grade | Parameter |
| Pain at injection site | 0 | None |
| | 1 | Mild: Minor reaction to touch |
| | 2 | Moderate: Cries/protests on touch |
| | 3 | Severe: Cries when limb is moved/spontaneously painful |
| Redness at injection site | | Record greatest surface diameter in mm |
| Swelling at injection site | | Record greatest surface diameter in mm |
| Fever* | | Record temperature in °C |
| Irritability/Fussiness 0 | | Behaviour as usual |
| | 1 | Mild: Crying more than usual/no effect on normal activity |
| | 2 | Moderate: Crying more than usual/interferes with normal activit |
| 3 | | Severe: Crying that cannot be comforted/prevents normal |
| | | activity |
| Drowsiness | 0 | Behaviour as usual |
| | 1 | Mild: Drowsiness easily tolerated |
| | 2 | Moderate: Drowsiness that interferes with normal activity |
| | 3 | Severe: Drowsiness that prevents normal activity |
| Loss of appetite | 0 | Appetite as usual |
| | 1 | Mild: Eating less than usual/no effect on normal activity |
| | 2 | Moderate: Eating less than usual/interferes with normal activity |
| | 3 | Severe: Not eating at all |

<sup>\*</sup> Fever is defined as temperature ≥ 38.0°C. The preferred location for measuring temperature in this study will be the axilla.

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

Table 7 Intensity scales for solicited symptoms in adults and children of six years of age or more

| | Adult/Chile | d (≥6 years) |
|---|---|---|
| Adverse Event | Intensity grade | Parameter |
| Pain at injection site | 0 | None |
| | 1 | Mild: Any pain neither interfering with nor preventing normal every day activities. |
| | 2 | Moderate: Painful when limb is moved and interferes with every day activities. |
| | 3 | Severe: Significant pain at rest. Prevents normal every day activities. |
| Redness at injection site | | Record greatest surface diameter in mm |
| Swelling at injection site | | Record greatest surface diameter in mm |
| Fever* | | Record temperature in °C |
| Headache | 0 | Normal |
| | 1 | Mild: Headache that is easily tolerated |
| | 2 | Moderate: Headache that interferes with normal activity |
| | 3 | Severe: Headache that prevents normal activity |
| Fatigue | 0 | Normal |
| | 1 | Mild: Fatigue that is easily tolerated |
| | 2 | Moderate: Fatigue that interferes with normal activity |
| Γ | 3 | Severe: Fatigue that prevents normal activity |
| Gastrointestinal symptoms | 0 | Normal |
| (nausea, vomiting, diarrhoea and/or abdominal pain) | 1 | Mild: Gastrointestinal symptoms that are easily tolerated |
| | 2 | Moderate: Gastrointestinal symptoms that interfere with normal activity |
| | 3 | Severe: Gastrointestinal symptoms that prevent normal activity |

<sup>\*</sup> Fever is defined as temperature  $\geq$  38.0°C. The preferred location for measuring temperature in this study will be the axilla.

The maximum intensity of local injection site redness/swelling for toddlers and children <6 years of age will be scored at GSK Biologicals as follows:

| 0 | Absent |
|---|------------------|
| 1 | ≤5 mm |
| 2 | >5 mm and ≤20 mm |
| 3 | >20 mm |

The maximum intensity of local injection site redness/swelling for adults and children ≥6 years of age will be scored at GSK Biologicals as follows:

| 0 | Absent |
|---|-------------------|
| 1 | ≤20 mm |
| 2 | >20 mm and ≤50 mm |
| 3 | >50 mm |

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

The maximum intensity of fever will be scored at GSK Biologicals as follows:

| 0 | <38℃ |
|---|----------------------|
| 1 | ≥38.0 °C to ≤39.0 °C |
| 2 | >39.0 °C to ≤40.0 °C |
| 3 | >40.0℃ |

Note that for all tables described in this section, the way the percentage of subjects will be derived will depend on the event analysed (see table below for details). As a result, the N value will differ from one table to another.

| Event | N used for deriving % per subject for<br>Vaccination phase | N used for deriving % per dose for<br>Vaccination phase |
|---|---|---|
| Concomitant vaccination | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Solicited general symptom | All subjects with solicited symptoms documented as present or absent for at least one dose. | All doses with solicited symptoms documented as present or absent within 0-3 days post dose |
| Unsolicited symptom | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Concomitant medication | All subjects with study vaccine administered | All study visits with study vaccine administered |

For summaries by MedDRA primary preferred term combining solicited and unsolicited adverse events, solicited adverse events will be coded as per the following MedDRA codes

| Solicited symptom | Lower level term code | Corresponding Lower level term decode |
|---|---|---|
| Headache | 10019211 | Drowsiness |
| Fatigue | 10016256 | Fatigue |
| Gastrointestinal symptoms | 10017944 | |
| Drowsiness | 10013649 | Drowsiness |
| Fever | 10016558 | Fever |
| Irritability/Fussiness | 10022998 | Irritability |
| Loss of appetite | 10003028 | Appetite lost |
| Pain at injection site | 10022086 | Injection site pain |
| Redness at injection site | 10022098 | Redness at injection site |
| Swelling at injection site | 10053425 | Swelling at injection site |

# 12. ANNEX 2: SUMMARY ON ELIMINATION CODES

Refer to section 5.2

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

# 13. ANNEX 3: STUDY SPECIFIC MOCK TFL

The following draft study specific mock TFLs will be used.

The data display, title and footnote are for illustration purpose and will be adapted to the study specificity such as one group and one dose for the study.

These templates were copied from recent studies. Note that there may be few changes between the study specific SAP mock TFL and the final TFLs. These editorial/minor changes will not lead to a SAP amendment.

Template 1 Number of subjects enrolled by center (Total Vaccinated Cohort)

| | Combo group | Control group | Total | |
|--------|-------------|---------------|-------|------|
| Center | n | N | n | % |
| PPD | 20 | 21 | 41 | 9.1 |
| PPD | 27 | 28 | 55 | 12.2 |
| PPD | 7 | 7 | 14 | 3.1 |
| PPD | 16 | 16 | 32 | 7.1 |
| PPD | 27 | 26 | 53 | 11.8 |
| PPD | 26 | 26 | 52 | 11.5 |
| PPD | 25 | 25 | 50 | 11.1 |
| PPD | 23 | 24 | 47 | 10.4 |
| PPD | 22 | 22 | 44 | 9.8 |
| PPD | 24 | 25 | 49 | 10.9 |
| PPD | 7 | 7 | 14 | 3.1 |
| All | 224 | 227 | 451 | 100 |

<sup>&</sup>lt;group description >

n = number of subjects included in each group or in total for a given center or for all centers

All = sum of all subjects in each group or in total (sum of all groups)

 $% = n/AII \times 100$ 

Template 2 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal at Visit 3 (Total Vaccinated Cohort)

| | HRV Liq | HRV<br>LYO | Total |
|---|---|---|---|
| Number of subjects vaccinated | 300 | 300 | 1200 |
| Number of subjects completed | 298 | 297 | 1193 |
| Number of subjects withdrawn | 2 | 3 | 7 |
| Reasons for withdrawal : | | | |
| Serious Adverse Event | 0 | 1 | 1 |
| Non-serious adverse event | 0 | 0 | 0 |
| Protocol violation | 0 | 0 | 0 |
| Consent withdrawal (not due to an adverse event) | 1 | 2 | 4 |
| Migrated/moved from study area | 1 | 0 | 2 |
| Lost to follow-up (subjects with incomplete vaccination course) | 0 | 0 | 0 |
| Lost to follow-up (subjects with complete vaccination course) | 0 | 0 | 0 |
| Others | 0 | 0 | 0 |

HRV LIQ = HRV vaccine liquid formulation

HRV LYO = HRV vaccine HRV Lyophilised formulation

Vaccinated = number of subjects who were vaccinated in the study

Completed = number of subjects who completed study visit 3

Withdrawn = number of subjects who did not come for study visit 3

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

# Template 3 Number of subjects at each visit and list of withdrawn subjects (Total Vaccinated Cohort)

| Group | VISIT | N | Withdrawn<br>Subject numbers | Reason for withdrawal |
|---|---|---|---|---|
| HRV Liq | VISIT 1 | 508 | | |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no PP | CONSENT WITHDRAWAL |
| | | | uo. PhD | CONSENT WITHDRAWAL |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 2 | 504 | | |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | SERIOUS ADVERSE EXPERIENCE |
| | VISIT 3 | 501 | | |
| | | | no. P | MIGRATION FROM STUDY AREA |
| | | | | CONSENT WITHDRAWAL |
| | | | no. Pr | MIGRATION FROM STUDY AREA |
| | | | no. Pr | CONSENT WITHDRAWAL |
| | | | no. Pr | MIGRATION FROM STUDY AREA |
| | | | no. Pr | MIGRATION FROM STUDY AREA |
| | | | no. Pru | CONSENT WITHDRAWAL |
| | | | no. PPD | MIGRATION FROM STUDY AREA |
| | | | no. PPD | MIGRATION FROM STUDY AREA |
| | VISIT 4 | 492 | | |
| HRV Lyo | VISIT 1 | 257 | | |
| , | | | no. PP | PROTOCOL VIOLATION |
| | | | uo. PhD | CONSENT WITHDRAWAL |
| | VISIT 2 | 255 | | |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 3 | 254 | | |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. Pr | LOST TO FOLLOW-UP |
| | | | no. Pr | LOST TO FOLLOW-UP |
| | | | no. Pr | CONSENT WITHDRAWAL |
| | | | no. Pr | MIGRATION FROM STUDY AREA |
| | | | no. Pru | LOST TO FOLLOW-UP |
| | | | no. PPD | ADVERSE EXPERIENCE |
| | VISIT 4 | 247 | | |

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

Template 4 Number of subjects enrolled into the study as well as the number of subjects excluded from ATP analyses with reasons for exclusion

| | | To | otal | | HRV LIQ | | | HRV LYO | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Title | N | n | S | % | N | n | S | N | n | S |
| Total enrolled cohort | 1200 | | | | 300 | | | 300 | | |
| TVC | 1200 | | | 100 | 300 | | | 300 | | |
| Administration of vaccine(s) forbidden in the | | 2 | 2 | | | 0 | 0 | | 0 | 0 |
| protocol | | | | | | | | | | |
| (code 1040) | | | | | | | | | | |
| Study vaccine dose not administered | | 73 | 73 | | | 23 | 23 | | 16 | 16 |
| according to protocol (code 1070) | | | | | | | | | | |
| Initially seropositive or unknown anti- | | 10 | 11 | | | 3 | 3 | | 1 | 1 |
| rotavirus IgA antibody on day of dose 1 | | | | | | | | | | |
| (code 1500) | | | | | | | | | | |
| Protocol violation (inclusion/exclusion | | 1 | 1 | | | 1 | 1 | | 0 | 0 |
| criteria) | | | | | | | | | | |
| (code 2010) | | | | | | | | | | |
| Administration of any medication forbidden | | 1 | 1 | | | 0 | 0 | | 1 | 1 |
| by the protocol (code 2040) | | | | | | | | | | |
| Underlying medical condition forbidden by | | 1 | 1 | | | 0 | 0 | | 0 | 0 |
| the protocol | | | | | | | | | | |
| (code 2050) | | | | | | | | | | |
| Concomitant infection not related to the | | 0 | 1 | | | 0 | 0 | | 0 | 1 |
| vaccine which may influence immune | | | | | | | | | | |
| response (code 2070) | | | | | | | | | | |
| Non compliance with vaccination schedule | | 14 | 16 | | | 6 | 7 | | 3 | 4 |
| (including wrong and unknown dates ) | | | | | | | | | | |
| (code 2080) | | | | | | | | | | |
| Non compliance with blood sampling | | 12 | 16 | | | 3 | 5 | | 4 | 5 |
| schedule (including wrong and unknown | | | | | | | | | | |
| dates) | | | | | | | | | | |
| (code 2090) | | | | | | | | | | |
| Essential serological data missing (code | | 87 | 95 | | | 20 | 22 | | 23 | 26 |
| 2100) | | | | | | | | | | |
| Subjects with incomplete study vaccination | | 1 | 1 | | | 0 | 0 | | 0 | 0 |
| schedule but with post serological result | | | | | | | | | | |
| (code 2500) | | | | | | | | | | $\perp$ |
| ATP | 998 | | | 83.2 | 244 | | | 252 | | $\perp$ |

HRV LIQ = HRV vaccine liquid formulation Lot C HRV LYO = HRV vaccine HRV Lyophilised formulation

Note: Subjects may have more than one elimination code assigned

n = number of subjects with the elimination code assigned excluding subjects who have been assigned a lower elimination code number

s = number of subjects with the elimination code assigned

<sup>% =</sup> percentage of subjects in the per protocol set (ATP) relative to the TVC (ES)

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

Template 5 Deviations from specifications for age and intervals between study visits (Total Vaccinated Cohort)

| | | Age | VA | AC_1-SER_2 |
|---|---|---|---|---|
| Group | | Protocol | Protocol | Adapted |
| - | | from 10 to 15 year | from 30 to 48 days | from 21 to 48 days |
| dTpaNew Group | N | 335 | 329 | 329 |
| | n | 0 | 11 | 8 |
| | % | 0.0 | 3.3 | 2.4 |
| | range | 10 to 15 | 28 to 74 | 28 to 74 |
| dTpaPre Group | N | 336 | 329 | 329 |
| | n | 0 | 10 | 8 |
| | % | 0.0 | 3.0 | 2.4 |
| | range | 10 to 15 | 29 to 95 | 29 to 95 |

HRV LIQ = HRV vaccine liquid formulation Lot A

HRV LIQ = HRV vaccine liquid formulation Lot B

HRV LIQ = HRV vaccine liquid formulation Lot C

HRV LYO = HRV vaccine HRV Lyophilised formulation

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

Adapted = interval used for defining the ATP cohorts for immunogenicity

N = total number of subjects with available results

n(%) = number(percentage) of subjects with results outside of the interval

range = minimum-maximum for age and intervals

VAC = vaccination

SER = Blood Sampling

Template 6 Summary of demographic characteristics (ATP cohort for Immunogenicity)

| | | dTpaNe<br>Group<br>N = 33 | ) | dTpaP<br>Grou<br>N = 33 | р | Tota<br>N = 67 | - |
|---|---|---|---|---|---|---|---|
| Characteristics | Parameters or Categories | Value or n | % | Value or n | % | Value or n | % |
| Age (years) at vaccination dose: 1 | Mean | 11.9 | - | 11.9 | - | 11.9 | - |
| | SD | 1.59 | - | 1.61 | - | 1.60 | - |
| | Median | 12.0 | - | 12.0 | - | 12.0 | - |
| | Minimum | 10 | - | 10 | - | 10 | - |
| | Maximum | 15 | - | 15 | - | 15 | - |
| Gender | Female | 179 | 53.4 | 178 | 53.0 | 357 | 53.2 |
| | Male | 156 | 46.6 | 158 | 47.0 | 314 | 46.8 |
| Geographic Ancestry | African Heritage / African American | 1 | 0.3 | 1 | 0.3 | 2 | 0.3 |
| | American Indian or Alaskan Native | 146 | 43.6 | 149 | 44.3 | 295 | 44.0 |
| | White - Arabic / North African<br>Heritage | 1 | 0.3 | 0 | 0.0 | 1 | 0.1 |
| | White - Caucasian / European<br>Heritage | 9 | 2.7 | 12 | 3.6 | 21 | 3.1 |
| | Other (Hispanic) | 178 | 53.1 | 174 | 51.8 | 352 | 52.5 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

N = total number of subjects

n(%) = Number(percentage) of subjects in a given category

Value = value of the considered parameter

SD = standard deviation

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

# Template 7 Summary of vital signs characteristics (Total Vaccinated Cohort)

| | | dTpaNew Group<br>(N = 335) | dTpaPre Group<br>(N = 336) | Total<br>(N = 671) |
|---|---|---|---|---|
| Characteristics | Parameters | Value | Value | Value |
| Height (km) | Mean | 152.6 | 151.5 | 152.1 |
| . , | SD | 10.48 | 10.44 | 10.47 |
| | Median | 152.0 | 151.5 | 152.0 |
| | Minimum | 112.0 | 126.0 | 112.0 |
| | Maximum | 189.0 | 187.0 | 189.0 |
| | Unknown | 0 | 0 | 0 |
| Weight (kg) | Mean | 49.7 | 48.8 | 49.2 |
| | SD | 13.23 | 13.61 | 13.42 |
| | Median | 47.0 | 47.1 | 47.0 |
| | Minimum | 28.0 | 19.4 | 19.4 |
| | Maximum | 99.0 | 110.0 | 110.0 |
| | Unknown | 0 | 0 | 0 |
| BMI (kg/m²) | Mean | 21.1 | 20.9 | 21.0 |
| , , | SD | 3.92 | 3.91 | 3.92 |
| | Median | 20.6 | 20.4 | 20.4 |
| | Minimum | 11.9 | 9.8 | 9.8 |
| | Maximum | 33.5 | 34.0 | 34.0 |
| | Unknown | 0 | 0 | 0 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

N = total number of subjects

Value = value of the considered parameter

SD = standard deviation

Height (cm) = Height expressed in centimeters

Weight (kg) = Weight expressed in kilograms

BMI (kg/m<sup>2</sup>) = Body Mass Index expressed in kilograms per meter square

# Template 8 Study population (Total Vaccinated Cohort)

| Number of subjects | Combo<br>group | Control group |
|---|---|---|
| Planned, N | 225 | 225 |
| Randomised, N (Total Vaccinated Cohort) | 224 | 227 |
| Completed, n (%) | 224 (100) | 227 (100) |
| Demographics | Combo | Control |
| | group | group |
| N (Total Vaccinated Cohort) | 224 | 227 |
| Females :Males | 97:127 | 115:112 |
| Mean Age, weeks (SD) | 8.8 (1.1) | 8.8 (1.1) |
| Median Age, weeks (minimum, maximum) | 9 (7, 11) | 9 (7, 11) |
| Most frequent race: Asian - East Asian Heritage, n (%) | 224 (100) | 226 (99.6) |

Combo group = Subjects received DTPa-IPV/Hib vaccine as a single injection at 2, 4 and 6 months of age

Control group = Subjects received DTPa-IPV and Hib vaccines at different injection sites at 2, 4 and 6 months of age

N = Total number of subjects enrolled in the study

n/% = Number/percentage of subjects in a given category

SD = Standard Deviation

MeaAge = Age calculated from Date of birth to first study vaccination

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

Template 9 Seropositivity and seroprotection rates and GMCs for anti-diphtheria and anti-tetanus antibodies before and one month after the booster vaccination (ATP cohort for immunogenicity)

| | | | | ≥ | assay | / cut- | off* | ≥ 0.1 IU/mL | | | | GMC | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95% | 6 CI | | | 95% | 6 CI | | | 6 CI |
| Antibody | Group | Timing | N | n | % | LL | UL | n | % | LL | UL | value | LL | UL |
| anti-diphtheria | dTpaNew Group | PRE | 321 | 284 | 88.5 | 84.5 | 91.8 | 83 | 25.9 | 21.2 | 31.0 | 0.472 | 0.403 | 0.553 |
| | | POST | 321 | 320 | 99.7 | 98.3 | 100 | 315 | 98.1 | 96.0 | 99.3 | 6.784 | 6.178 | 7.450 |
| | dTpaPre Group | PRE | 319 | 286 | 89.7 | 85.8 | 92.8 | 89 | 27.9 | 23.0 | 33.2 | 0.456 | 0.392 | 0.530 |
| | | POST | 319 | 319 | 100 | 98.9 | 100 | 310 | 97.2 | 94.7 | 98.7 | 6.493 | 5.915 | 7.128 |
| anti-tetanus | dTpaNew Group | PRE | 321 | 311 | 96.9 | 94.3 | 98.5 | 151 | 47.0 | 41.5 | 52.7 | 0.956 | 0.835 | 1.095 |
| | | POST | 321 | 321 | 100 | 98.9 | 100 | 321 | 100 | 98.9 | 100 | 18.937 | 17.313 | 20.713 |
| | dTpaPre Group | PRE | 319 | 314 | 98.4 | 96.4 | 99.5 | 143 | 44.8 | 39.3 | 50.5 | 0.899 | 0.789 | 1.026 |
| | | POST | 319 | 319 | 100 | 98.9 | 100 | 319 | 100 | 98.9 | 100 | 18.515 | 16.851 | 20.342 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

Seroprotection=anti-diphtheria and anti-tetanus antibody concentration ≥0.1 IU/mL

\*Assay cut-off is 0.057 IU/mL and 0.043 IU/mL for anti-diphtheria and anti-tetanus respectively

GMC = geometric mean antibody concentration calculated on all subjects

N = number of subjects with available results

n(%)=number(percentage) of subjects with antibody concentrations above the specified cut-off

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

PRE=Pre-booster blood sampling time point

POST=Post-booster blood sampling time point

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

Template 10 Booster responses for anti-PT, anti-FHA and anti-PRN antibody concentration one month after the booster vaccination (ATP cohort for immunogenicity)

| | | | | | Booste | r respo | ıse |
|---|---|---|---|---|---|---|---|
| | | | | | | | 5% CI |
| anti-FHA | Group | Pre-vaccination status | N | n | % | LL | UL |
| anti-PT | dTpaNew Group | S- | 142 | 135 | 95.1 | 90.1 | 98.0 |
| | | S+ (< 4*assay cut-off) | 104 | 103 | 99.0 | 94.8 | 100 |
| | | S+ (≥4*assay cut-off) | 71 | 60 | 84.5 | 74.0 | 92.0 |
| | | Total | 317 | 298 | 94.0 | 90.8 | 96.4 |
| | dTpaPre Group | S- | 143 | 131 | 91.6 | 85.8 | 95.6 |
| | | S+ (<4*assay cut-off) | 114 | 112 | 98.2 | 93.8 | 99.8 |
| | | S+ (≥4*assay cut-off) | 61 | 52 | 85.2 | 73.8 | 93.0 |
| | | Total | 318 | 295 | 92.8 | 89.3 | 95.4 |
| anti-FHA | dTpaNew Group | S- | 6 | 6 | 100 | 54.1 | 100 |
| | | S+ (<4*assay cut-off) | 57 | 57 | 100 | 93.7 | 100 |
| | | S+ (≥4*assay cut-off) | 251 | 242 | 96.4 | 93.3 | 98.3 |
| | | Total | 314 | 305 | 97.1 | 94.6 | 98.7 |
| | dTpaPre Group | S- | 5 | 5 | 100 | 47.8 | 100 |
| | | S+ (<4*assay cut-off) | 55 | 55 | 100 | 93.5 | 100 |
| | | S+ (≥4*assay cut-off) | 255 | 244 | 95.7 | 92.4 | 97.8 |
| | | Total | 315 | 304 | 96.5 | 93.8 | 98.2 |
| anti-PRN | dTpaNew Group | S- | 52 | 50 | 96.2 | 86.8 | 99.5 |
| | | S+ (<4*assay cut-off) | 152 | 151 | 99.3 | 96.4 | 100 |
| | | S+ (≥4*assay cut-off) | 117 | 114 | 97.4 | 92.7 | 99.5 |
| | | Total | 321 | 315 | 98.1 | 96.0 | 99.3 |
| | dTpaPre Group | S- | 47 | 47 | 100 | 92.5 | 100 |
| | | S+ (<4*assay cut-off) | 159 | 159 | 100 | 97.7 | 100 |
| | | S+ (≥4*assay cut-off) | 112 | 111 | 99.1 | 95.1 | 100 |
| | | Total | 318 | 317 | 99.7 | 98.3 | 100 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

Total = subjects either seropositive or seronegative at pre-vaccination

S- = seronegative subjects (antibody concentration below assay cut off for anti-PT, anti-FHA, anti-PRN)

S+ = seropositive (antibody concentration below assay cut off for anti-PT, anti-FHA, anti-PRN)

Booster response to PT, FHA and PRN antigens is defined as:

- initially seronegative subjects (pre-booster antibody concentration below the assay cut-off) with an increase
  of at least four times the assay cut-off one month after vaccination.
- initially seropositive subjects with anti-body concentration < four times the assay cut-off with an increase of at least four times the pre-booster antibody concentration one month after vaccination
- initially seropositive subjects with anti-body concentration ≥ four times the assay cut-off with an increase of at least two times the pre-booster antibody concentration one month after vaccination

Assay cut-off is 2.693 IU/mL, 2.046 IU/mL and 2.187 IU/mL for anti-PT, FHA and PRN respectively

N = number of subjects with both pre- and post-vaccination results available

n(%) = number(percentage) of subjects with a booster response

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

S- = Initially seronegative subjects prior to vaccination

S+ = Initially seropositive subjects prior to vaccination

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

Template 11 Reverse cumulative curve for anti-diphtheria antibody concentration one month after the booster vaccination (ATP cohort for immunogenicity)



dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

# Template 12 Seroprotection rate for anti-Diphtheria antibody concentration by ELISA and VERO NEUTRALISATION (ATP cohort)

| | | | conce | LISA<br>entrations<br>w the 0.1<br>U/ml | below<br>among<br>ELISA | among subjects with | | Neutra<br>concentrations below<br>the 0.01 IU/ml among<br>subjects with ELISA<br>results | | | ted<br>on of<br>ubjects<br>s 95% |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Group | Timing | N | n/N | % | n'/N' | % | n/N x n'/N' | % | SP | LL | UL |
| (each group) | Pre | | | | | | | | | | |
| 5 17 | post | | | | | | | | | | |

Boostrix group= Subjects who had received GSK Biologicals' Tdap vaccine (Boostrix) in study 106316 and a second dose of Tdap vaccine (Boostrix) at Year 9 Visit 6

Adacel group= Subjects who had received Sanofi Pasteurs' Tdap vaccine (Adacel) in study 106316 and a second dose of Tdap vaccine (Boostrix) at Year 9 Visit 6

N = number of subjects tested by ELISA

N' = number of subjects with ELISA concentrations below the 0.1 IU/ml who were tested by Vero

% = proportion of subjects with concentrations below the considered cut-off (0.1 IU/ml for ELISA and 0.01 IU/ml for

VERO) n/N x n'/N' = the multiplication of the two proportions = overall seronegativity for anti-Diphtheria

Overall = based on both the ELISA and the Vero-cell neutralisation testing

95% CI = exact 95% confidence interval; LL = lower limit, UL = upper limit

Pre= blood sampling, at Month 0 before vaccination

post= blood sampling, one moth after vaccination

SP= proportion of subjects with either ELISA concentrations above 0.1 IU/ml or Neutra concentration above 0.01 IU/mL

Template 13 Compliance in returning symptom information (Total Vaccinated Cohort)

| Group | Number<br>of<br>doses | Doses NOT according to protocol | Number<br>of<br>general SS | Compliance<br>%<br>general SS | Number<br>of<br>local SS | Compliance<br>%<br>local SS |
|---|---|---|---|---|---|---|
| dTpaNew Group | 335 | 0 | 330 | 98.5 | 330 | 98.5 |
| dTpaPre Group | 336 | 1 | 329 | 97.9 | 329 | 97.9 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

SS = Symptom screens/sheets used for the collection of local and general solicited AEs

Compliance % = (number of doses with symptom screen/sheet return / number of administered doses) X 100

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

Template 14 Incidence and nature of grade 3 symptoms (solicited and unsolicited) reported during the 4-day (Days 0-3) period after vaccination following each dose and overall (Total Vaccinated Cohort)

| | | An | y sym | ptom | | General symptoms | | | | | Local symptoms | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% | 6 CI | | 95% | | | | | | | 95% CI | |
| Group | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| dTpaNew Group | 335 | 264 | 78.8 | 74.0 | 83.1 | 335 | 134 | 40.0 | 34.7 | 45.5 | 335 | 250 | 74.6 | 69.6 | 79.2 |
| dTpaPre Group | 336 | 279 | 83.0 | 78.6 | 86.9 | 336 | 151 | 44.9 | 39.5 | 50.4 | 336 | 264 | 78.6 | 73.8 | 82.8 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

n(%)= number(percentage) of subjects presenting at least one type of symptom whatever the study vaccine administered

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Template 15 Incidence of solicited local symptoms reported during the 4-day (Days 0-3) period after vaccination following each dose and overall (Total Vaccinated Cohort)

| | | | dΤ | paNew | Group | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 | % CI | | | | 95 | % CI |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL |
| Pain | All | 330 | 237 | 71.8 | 66.6 | 76.6 | 329 | 248 | 75.4 | 70.4 | 79.9 |
| | Grade 3 | 330 | 24 | 7.3 | 4.7 | 10.6 | 329 | 20 | 6.1 | 3.8 | 9.2 |
| | Medical advice | 330 | 0 | 0.0 | 0.0 | 1.1 | 329 | 0 | 0.0 | 0.0 | 1.1 |
| Redness (mm) | All | 330 | 113 | 34.2 | 29.1 | 39.6 | 329 | 94 | 28.6 | 23.8 | 33.8 |
| | Grade 3 | 330 | 4 | 1.2 | 0.3 | 3.1 | 329 | 1 | 0.3 | 0.0 | 1.7 |
| | Medical advice | 330 | 0 | 0.0 | 0.0 | 1.1 | 329 | 0 | 0.0 | 0.0 | 1.1 |
| Swelling (mm) | All | 330 | 98 | 29.7 | 24.8 | 34.9 | 329 | 90 | 27.4 | 22.6 | 32.5 |
| - ' ' | Grade 3 | 330 | 6 | 1.8 | 0.7 | 3.9 | 329 | 5 | 1.5 | 0.5 | 3.5 |
| | Medical advice | 330 | 0 | 0.0 | 0.0 | 1.1 | 329 | 0 | 0.0 | 0.0 | 1.1 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

N = number of subjects with the administered dose

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

N = number of subjects with the documented dose

n(%)= number(percentage) of subjects reporting the symptom at least once

<sup>95%</sup>CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

# Template 16 Incidence of solicited general symptoms reported during the 4-day (Days 0-3) post-vaccination period (Total Vaccinated Cohort)

| | | | dΤι | paNew | Grou | р | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 | % CI | | - | | 95 | % CI |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL |
| Fatigue | All | 330 | 83 | 25.2 | 20.6 | 30.2 | 329 | 86 | 26.1 | 21.5 | 31.2 |
| | Grade 3 | 330 | 7 | 2.1 | 0.9 | 4.3 | 329 | 4 | 1.2 | 0.3 | 3.1 |
| | Related | 330 | 77 | 23.3 | 18.9 | 28.3 | 329 | 83 | 25.2 | 20.6 | 30.3 |
| | Medical advice | 330 | 1 | 0.3 | 0.0 | 1.7 | 329 | 1 | 0.3 | 0.0 | 1.7 |
| Gastrointestinal | All | 330 | 32 | 9.7 | 6.7 | 13.4 | 329 | 42 | 12.8 | 9.4 | 16.9 |
| | Grade 3 | 330 | 3 | 0.9 | 0.2 | 2.6 | 329 | 3 | 0.9 | 0.2 | 2.6 |
| | Related | 330 | 29 | 8.8 | 6.0 | 12.4 | 329 | 40 | 12.2 | 8.8 | 16.2 |
| | Medical advice | 330 | 2 | 0.6 | 0.1 | 2.2 | 329 | 1 | 0.3 | 0.0 | 1.7 |
| Headache | All | 330 | 88 | 26.7 | 22.0 | 31.8 | 329 | 108 | 32.8 | 27.8 | 38.2 |
| | Grade 3 | 330 | 5 | 1.5 | 0.5 | 3.5 | 329 | 3 | 0.9 | 0.2 | 2.6 |
| | Related | 330 | 80 | 24.2 | 19.7 | 29.2 | 329 | 103 | 31.3 | 26.3 | 36.6 |
| | Medical advice | 330 | 2 | 0.6 | 0.1 | 2.2 | 329 | 1 | 0.3 | 0.0 | 1.7 |
| Temperature/(Axillary) (°C) | All | 330 | 9 | 2.7 | 1.3 | 5.1 | 329 | 6 | 1.8 | 0.7 | 3.9 |
| | ≥37.5 | 330 | 9 | 2.7 | 1.3 | 5.1 | 329 | 6 | 1.8 | 0.7 | 3.9 |
| | >38.0 | 330 | 5 | 1.5 | 0.5 | 3.5 | 329 | 1 | 0.3 | 0.0 | 1.7 |
| | >38.5 | 330 | 3 | 0.9 | 0.2 | 2.6 | 329 | 1 | 0.3 | 0.0 | 1.7 |
| | >39.0 | 330 | 2 | 0.6 | 0.1 | 2.2 | 329 | 0 | 0.0 | 0.0 | 1.1 |
| | Related | 330 | 7 | 2.1 | 0.9 | 4.3 | 329 | 6 | 1.8 | 0.7 | 3.9 |
| | Medical advice | 330 | 2 | 0.6 | 0.1 | 2.2 | 329 | 0 | 0.0 | 0.0 | 1.1 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

N = number of subjects with the documented dose

n(%)= number(percentage) of subjects reporting the symptom at least once

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

Related = Symptoms which is assessed by the investigator as related to vaccination

Grade3\*Related = Grade 3 symptom which is assessed by the investigator as related to vaccination

Grade 3 For Headache: Headache that prevented normal activity

For Fatigue: Fatigue that prevented normal activity

For Gastrointestinal symptoms: Gastrointestinal symptoms that prevented normal activity

For Fever: >39.0 °C

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

Template 17 Percentage of subjects with grade 3 unsolicited symptoms classified by MedDRA SOC and PT from Day 0 to Day 30 after any vaccination (Total Vaccinated Cohort)

| Primary System Organ | Preferred | | | LIQ<br>298 | | | | / LIQ<br>: 302 | | | | / LIQ<br>300 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Class (CODE) | Term (CODE) | | | 95% | 6 CI | | | 95 | % CI | | | 95 | % CI |
| , | , | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| At least one symptom | | 24 | 8.1 | 5.2 | 11.7 | 26 | 8.6 | 5.7 | 12.4 | 33 | 11.0 | 7.7 | 15.1 |
| Ear and labyrinth | Ear pain | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| disorders (10013993) | (10014020) | | | | | | | | | | | | |
| Eye disorders (10015919) | Conjunctivitis (10010741) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 1 | 0.3 | 0.0 | 1.8 |
| Gastrointestinal disorders (10017947) | Diarrhoea<br>(10012735) | 0 | 0.0 | 0.0 | 1.2 | 2 | 0.7 | 0.1 | 2.4 | 1 | 0.3 | 0.0 | 1.8 |
| , | Flatulence (10016766) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 2 | 0.7 | 0.1 | 2.4 |
| General disorders and administration site conditions (10018065) | Injection site erythema (10022061) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| , | Injection site pain (10022086) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Injection site<br>swelling<br>(10053425) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Irritability<br>(10022998) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 1 | 0.3 | 0.0 | 1.8 |
| | Pyrexia (10037660) | 4 | 1.3 | 0.4 | 3.4 | 3 | 1.0 | 0.2 | 2.9 | 4 | 1.3 | 0.4 | 3.4 |
| Immune system disorders (10021428) | Hypersensitivit y (10020751) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| Infections and infestations (10021881) | Bronchitis<br>(10006451) | 2 | 0.7 | 0.1 | 2.4 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| , | Ear infection<br>(10014011) | 1 | 0.3 | 0.0 | 1.9 | 3 | 1.0 | 0.2 | 2.9 | 2 | 0.7 | 0.1 | 2.4 |
| | Exanthema subitum (10015586) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| | Eye infection (10015929) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Gastroenteritis (10017888) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Impetigo<br>(10021531) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Influenza<br>(10022000) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| | Laryngitis<br>(10023874) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Otitis media (10033078) | 5 | 1.7 | 0.5 | 3.9 | 6 | 2.0 | 0.7 | 4.3 | 11 | 3.7 | 1.8 | 6.5 |
| | Perianal<br>abscess<br>(10034447) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

| | | | | / LIQ | 1 Idii | | | HRV LIQ | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Primary System Organ | Preferred | | N = | 298 | | | N = | 302 | | | N = | 300 | |
| Class (CODE) | Term (CODE) | | | 95% | | | | 95 | % CI | | | 95 | % CI |
| | | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| | Pneumonia<br>(10035664) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| | Respiratory<br>tract infection<br>(10062352) | 3 | 1.0 | 0.2 | 2.9 | 2 | 0.7 | 0.1 | 2.4 | 0 | 0.0 | 0.0 | 1.2 |
| | Respiratory<br>tract infection<br>viral<br>(10062106) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Rhinitis<br>(10039083) | 2 | 0.7 | 0.1 | 2.4 | 1 | 0.3 | 0.0 | 1.8 | 3 | 1.0 | 0.2 | 2.9 |
| | Upper<br>respiratory tract<br>infection<br>(10046306) | 2 | 0.7 | 0.1 | 2.4 | 5 | 1.7 | 0.5 | 3.8 | 7 | 2.3 | 0.9 | 4.7 |
| | Varicella<br>(10046980) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 2 | 0.7 | 0.1 | 2.4 |
| Psychiatric disorders (10037175) | Crying (10011469) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| Respiratory, thoracic and mediastinal disorders (10038738) | Cough<br>(10011224) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 6 | 2.0 | 0.7 | 4.3 |
| | Nasal<br>congestion<br>(10028735) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Rales<br>(10037833) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| Skin and subcutaneous tissue disorders (10040785) | Dermatitis<br>allergic<br>(10012434) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| | Eczema<br>(10014184) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Rash<br>(10037844) | 2 | 0.7 | 0.1 | 2.4 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |

HRV LIQ = HRV vaccine liquid formulation Lot A HRV LIQ = HRV vaccine liquid formulation Lot B

HRV LIQ = HRV vaccine liquid formulation Lot C

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting at least once a specified unsolicited symptom

At least one symptom = number of subjects reporting at least one unsolicited symptom, whatever the MedDRA PT

95% CI = exact 95% Confidence Interval, LL = Lower Limit, UL = Upper Limit

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

# Template 18 Number (%) of subjects with serious adverse events from first study vaccination up to Visit 3 including number of events reported (Total Vaccinated Cohort)

| | | | | Gr 1<br>N = | | Gr2<br>N = | | |
|---|---|---|---|---|---|---|---|---|
| Type of Event | Primary System Organ<br>Class | Preferred Term (CODE) | n* | n | % | n* | n | % |
| SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Related SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Fatal SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Related fatal SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |

Gr 1 = Group 1 description

Gr 2 = Group 2 description

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

# Template 19 Subjects with Serious Adverse Events reported up to Visit 2 (Total Vaccinated Cohort)

| Sub.<br>No. | Case Id | Age at onset (Week) | Sex | Verbatim | Preferred term | System Organ<br>Class | MA<br>type | Dose | Day of onset | Duration | Causality | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| P | PPD | 12 | М | Kawasaki's<br>disease | Kawasaki's<br>disease | Infections and infestations | НО | 1 | 12 | 29 | N | Recovered/resolved |
| PP<br>D | PPD | 18 | М | Influenza-b | Influenza | Infections and infestations | НО | 2 | 2 | 5 | N | Recovered/resolved |
| PP<br>D | PPD | 17 | М | Acute gastroenteritis | Gastroenteritis | Infections and infestations | НО | 2 | 9 | 5 | N | Recovered/resolved |
| PP<br>D | PPD | 17 | F | Infantile spasms | Infantile spasms | Nervous system disorders | НО | 2 | 2 | 51 | N | Recovered/resolved with sequelae |
| PP<br>D | PPD | 21 | M | Rs-virus<br>bronchiolitis | Respiratory syncytial virus bronchiolitis | Infections and infestations | НО | 2 | 30 | 16 | N | Recovered/resolved |
| PP<br>D | PPD | 13 | М | Gastroenteritis | Gastroenteritis | Infections and infestations | НО | 1 | 25 | 6 | N | Recovered/resolved |
| PP<br>D | PPD | 22 | М | Pneumonia | Pneumonia | Infections and infestations | НО | 2 | 32 | 13 | N | Recovered/resolved |
| | | 23 | | Middle ear infection | Otitis media | Infections and infestations | НО | 2 | 37 | 8 | N | Recovered/resolved |
| PP<br>D | PPD | 14 | F | Secretory otitis media | Otitis media | Infections and infestations | НО | 1 | 7 | 25 | N | Recovered/resolved |
| PPD | PPD | 20 | М | Viral pneumonia | Pneumonia viral | Infections and infestations | НО | 2 | 13 | 23 | N | Recovered/resolved |
| PPD | PPD | 14 | М | Middle ear infection, left | Otitis media | Infections and infestations | НО | 1 | 19 | 8 | N | Recovered/resolved |
| | | 14 | | Pneumonia | Pneumonia | Infections and infestations | НО | 1 | 19 | 8 | N | Recovered/resolved |
| PPD | PPD | 13 | М | Acute lymphadenitis | Lymphadenitis | Blood and lymphatic system disorders | НО | 1 | 13 | 22 | N | Recovered/resolved |
| PPD | PPD | 10 | F | | Pyelonephritis acute | Infections and infestations | НО | 1 | 6 | 12 | N | Recovered/resolved |
| PPD | PPD | 19 | М | Laryngitis | Laryngitis | Infections and infestations | НО | 2 | 11 | 7 | N | Recovered/resolved |

# 201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

| Sub. | Case Id | Age at | Sex | Verbatim | Preferred term | System Organ | MA | Dose | Day of | Duration | Causality | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| No. | | onset<br>(Week) | | | | Class | type | | onset | | | |
| PPD | PPD | 14 | М | Bronchitis acuta | Bronchitis | Infections and infestations | НО | 1 | 23 | 12 | N | Recovered/resolved |
| | PPD | 19 | М | Bronchiolitis acuta | Bronchiolitis | Infections and infestations | НО | 2 | 26 | 7 | N | Recovered/resolved |
| | PPD | 19 | F | Laryngitis acuta | Laryngitis | Infections and infestations | НО | 2 | 7 | 4 | N | Recovered/resolved |
| PPD | PPD | 18 | F | Laryngitis | Laryngitis | Infections and infestations | НО | 2 | 7 | 4 | N | Recovered/resolved |
| PPD | PPD | 14 | F | Gastroenteritis | Gastroenteritis | Infections and infestations | НО | 1 | 22 | 7 | N | Recovered/resolved |

MA = medical attention

HO = hospitalisation

Dose = dose given prior to the start of the SAE
Day of onset = number of days since last study vaccine dose

Page 45 of 48 10-MAR-2019

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

Template 20 Number and percentage of subjects who started at least one concomitant medication from Day 0 to Day 7 (Total Vaccinated Cohort)

| | | ď | TpaNew | Group | | | dTpaPre Group | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 9 | 95% CI | | | 9 | 5% CI | |
| | N | n | % | LL | UL | N | n | % | LL | UL |
| Any | 335 | 41 | 12.2 | 8.9 | 16.2 | 336 | 43 | 12.8 | 9.4 | 16.8 |
| Any antipyretic | 335 | 37 | 11.0 | 7.9 | 14.9 | 336 | 41 | 12.2 | 8.9 | 16.2 |
| Prophylactic antipyretic | 335 | 2 | 0.6 | 0.1 | 2.1 | 336 | 2 | 0.6 | 0.1 | 2.1 |

dTpaNew Group = Subjects who received *Boostrix* in new syringe presentation

n(%)= number(percentage) of subjects who started to take the specified concomitant medication at least once during the mentioned period

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Template 21 Solicited and Unsolicited symptoms experienced by subjects classified by MedDRA Primary System Organ Class and Preferred Term within the 31-day (Days 0-30) post-vaccination period - SAE excluded (Total vaccinated cohort)

| | | HPV<br>N | MM | MMR_DTPa<br>N = | | | |
|---|---|---|---|---|---|---|---|
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n* | n | % | n* | n | % |
| At least one symptom | | | | | | | |
| <each soc=""></each> | <each pt="" term=""></each> | | | | | | |

HPV\_2D = females aged 4-6 years who received two doses of HPV-16/18 L1 VLP AS04 vaccine at Day 0 and Month 6 MMR\_DTPa = females aged 4-6 years who received MMR vaccine at Day 0 and DTPa vaccine at Month 6 At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n/% = number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Template 22 Minimum and maximum activity dates (TVC)

| Visit | Minimum date | Maximum date |
|-------|--------------|--------------|
| 1 | 19JUN2007 | 29DEC2007 |
| 2 | 24JUL2007 | 08FEB2008 |
| 3 | 24AUG2007 | 18MAR2008 |
| 4 | 25MAR2008 | 22NOV2008 |
| 5 | 24MAR2009 | 31MAR2009* |

<sup>\*</sup>Database Lock Date = 31MAR2009

dTpaPre Group = Subjects who received *Boostrix* in previous syringe presentation

N = number of subjects with the administered dose

n\* = number of events reported

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

# Template 23 Number of enrolled subjects by age category (TVC)

| | | Gr 1<br>N = | Gr 2<br>N = | Gr 3<br>N = | Total<br>N = |
|---|---|---|---|---|---|
| Characteristics | Categories | n | n | n | n |
| Age category | In utero | | | | |
| | Preterm newborn infants | | | | |
| | (gestational age < 37 wks) | | | | |
| | Newborns (0-27 days) | | | | |
| | Infants and toddlers (28 days- | | | | |
| | 23 months) | | | | |
| | Children (2-11 years) | | | | |
| | Adolescents (12-17 years) | | | | |
| | Adults (18-64 years) | | | | |
| | From 65-84 years | | | | |
| | 85 years and over | | | | |
| | Missing | | | | |

Gr 1 = Group 1 description

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories Missing = <describe missing>

# Template 24 Number of subjects by country

| | ACWY-TT | ACWYHPV | HPV | Co-ad | Tdap | Total |
|---|---|---|---|---|---|---|
| | N = 259 | N = 259 | N = 261 | N = 260 | N = 261 | N = 1300 |
| Country | n | n | N | n | n | n |
| Dominican Republic | 86 | 87 | 88 | 87 | 87 | 435 |
| Estonia | 87 | 86 | 87 | 87 | 88 | 435 |
| Thailand | 86 | 86 | 86 | 86 | 86 | 430 |

ACWY-TT = Subjects who received MenACWY-TT at Month 0 and Cervarix at Month 1, 2 and 7

ACWYHPV = Subjects who received MenACWY-TT and Cervarix at Month 0 and Cervarix at Month 1 and 6 HPV = Subjects who received Cervarix at Month 0. 1 and 6

HPV = Subjects who received Cervanx at Month U, I and 6

Co-ad = Subjects who received MenACWY-TT, Cervarix and Boostrix at Month 0 and Cervarix at Month 1 and 6 Tdap = Subjects who received Boostrix and Cervarix at Month 0 and Cervarix at Month 1 and 6 N = number of subjects

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories

# Template 25 Listing of dropouts due to AEs, SAEs and solicited symptoms (Total cohort)

| Study-<br>Subject<br>No. | Country | Gender | AE Description | SAE | Causality | Outcome | Type of discontinuation |
|---|---|---|---|---|---|---|---|
| PP<br>D | Germany | F | SUBJECT DIED | Υ | | Fatal | Study at visit/contact: VISIT11 (Y5) |
| PP<br>D | Germany | F | SUBJECT DIED | Υ | | Fatal | Study at visit/contact: VISIT11 (Y5) |

Gr 2 = Group 2 description

Gr 3 = Group 3 description

N = Number of enrolled subjects

201532 [DTPA (BOOSTRIX)-050] Statistical Analysis Plan Amendment 1 Final

# Template 26 Percentage of subjects with large injection site reaction during the 4-day (Days 0-3) period after Boostrix (Total Vaccinated Cohort)

| Type of Swelling | | (Each group)<br>N= | | | Total<br>N= | | |
|---|---|---|---|---|---|---|---|
| | n | n % 95%Cl | | | % | 95% CI | |
| | | | LL | UL | | LL | UL |
| Any | | | | | | | |
| Local Swelling | | | | | | | |
| Diffuse Swelling | | | | | | | |
| Involving at least one adjacent | | | | | | | |
| joint | | | | | | | |

Boostrix group= Subjects who had received GSK Biologicals' Tdap vaccine (Boostrix) in study 106316 and a second dose of Tdap vaccine (Boostrix) at Year 9 Visit 6

Adacel group= Subjects who had received Sanofi Pasteurs' Tdap vaccine (Adacel) in study 106316 and a second dose of Tdap vaccine (Boostrix) at Year 9 Visit 6

Control group= Subjects who will receive the first dose of Tdap vaccine (Boostrix) at Year 9 Visit 6

N = Number of subjects with documented dose

n/% = number/percentage of subjects reporting a specified symptom

95% CI = Standardized asymptotic 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Template 27 GMCs fold increase for anti-D, anti-T, anti-PT, anti-FHA and anti-PRN antibodies one month after the booster vaccination by study (Per protocol cohort for analysis of immunogenicity)

| | | | | | | | GN | C ratio | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | 95 | % |
| | | | | | | | | | C | ) |
| Antibody | Sub-grp | N | Time point | <b>GMC</b> | Time point | <b>GMC</b> | Ratio | Value | LL | UL |
| - | | | description | | description | | order | | | |
| Anti-Diphtheria | | | POST | | PRE | | POST / | | | |
| (IU/mL) | | | | | | | PRE | | | |

GMC = geometric mean antibody concentration

N = Number of subjects with available results at the two considered time points

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

PRE = blood sample taken before the booster vaccination

POST = blood sample taken one month after the booster vaccination